CLINICAL TRIAL: NCT03285763
Title: A Phase III/IV, Single Arm, Multicenter Study of Atezolizumab (Tecentriq) to Investigate Long-term Safety and Efficacy in Previously-treated Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer (TAIL)
Brief Title: A Study of Atezolizumab (Tecentriq) to Investigate Long-term Safety and Efficacy in Previously-treated Participants With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC)
Acronym: TAIL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO39171; 2017-001409-34 (EudraCT Number)
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab (Experimental): Participants with Stage IIIb or State IV NSCLC who have progressed after standard systemic chemotherapy will receive atezolizumab until Investigator-assessed loss of clinical benefit, unacceptable toxicity, investigator or participant's decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Participants will receive 1200 milligrams (mg) of atezolizumab administered by intravenous infusion on Day 1 of every 3-week cycle until Investigator-assessed loss of clinical benefit, unacceptable toxicity, investigator or participant's decision to withdraw from therapy, or death (whichever occurs first).
  Other Names: RO5541267; Tecentriq

SUMMARY:
This is a Phase III/IV, single-arm, multicenter study of the long-term safety and efficacy of atezolizumab treatment in participants with Stage IIIb or Stage IV NSCLC who have progressed after standard systemic chemotherapy (including if given in combination with anti-programmed cell death protein 1 [anti-PD-1] therapy, after anti-PD-1 as monotherapy, or after tyrosine kinase inhibitor [TKI] therapy). The study will consist of a Screening Period, a Treatment Period, a Treatment Discontinuation Visit, and a Follow-Up Period.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented Stage IIIb or Stage IV NSCLC that has progressed following standard systemic chemotherapy (including if given in combination with anti-PD-1 therapy, after anti-PD-1 as monotherapy, or after TKI therapy). Participants with a previously detected sensitizing epidermal growth factor receptor (EGFR) mutation or echinoderm microtubule-associated protein-like 4-anaplastic lymphoma kinase (ALK) fusion oncogene must have received targeted therapy (TKI) followed by at least one line of standard systemic chemotherapy prior to receiving atezolizumab. Overall, participants should not have received more than two lines of standard systemic chemotherapy. Participants who have discontinued first-line or second-line therapy due to intolerance are also eligible
* The last dose of prior systemic anticancer therapy or targeted therapy must have been administered more than or equal to (≥) 21 days prior to randomization.
* The last dose of prior anti-PD-1 therapy must have been administered. Nivolumab must have been discontinued >= 14 days and pembrolizumab >= 21 days prior to study treatment initiation, providing that these treatments were not administered in a clinical trial setting.
* Measurable disease, as defined by Response Evaluation Criteria for Solid Tumors, Version 1.1 (RECIST v1.1)
* Participants with asymptomatic central nervous system (CNS) metastases (treated or untreated), as determined by computed tomography (CT) or magnetic resonance imaging evaluation during screening and prior radiographic evaluation, are eligible
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Life expectancy ≥ 12 weeks
* Adequate hematologic and end-organ function
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of less than (<) 1 percent (%) per year during the treatment period and for at least 5 months after the last dose of atezolizumab
* Participants must have recovered (i.e., improvement to Grade 1 or better) from all acute toxicities from previous therapy, excluding alopecia and toxicities related to prior anti-PD-1-therapy

Exclusion Criteria:

* Symptomatic CNS metastases
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for ≥ 2 weeks prior to study treatment initiation
* Leptomeningeal disease
* Uncontrolled pericardial effusion or ascites requiring recurrent drainage procedures
* Pregnant or lactating, or intending to become pregnant during the study
* Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome)
* Significant cardiovascular disease, such as New York Heart Association cardiac disease ≥ Class III, myocardial infarction within 3 months, unstable arrhythmias, or unstable angina
* Significant renal disorder requiring dialysis or indication for renal transplant
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to study treatment initiation
* Major surgical procedure within 4 weeks prior to study treatment initiation or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis
* Inability to understand the local language(s) for which the EORTC QLQ-LC13 and EQ-5D-5L questionnaires are available
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* History of autoimmune disease are allowed if controlled and on stable treatment (i.e., same treatment, same dose) for the last 12 weeks
* Prior allogeneic stem cell or solid organ transplantation
* History of idiopathic pulmonary fibrosis, including pneumonitis, drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan
* Active tuberculosis
* Administration of a live, attenuated vaccine within 4 weeks prior to study treatment initiation
* Prior treatment with cluster of differentiation 137 (CD137) agonists or immune checkpoint blockade therapies other than anti-PD-1 therapy, including anti-programmed death-ligand 1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferons or interleukin-2) within 4 weeks or five half-lives of the drug, whichever is longer, prior to initiation of study treatment
* Specifically for participants without autoimmune disease: treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to study treatment initiation, or anticipated requirement for systemic immunosuppressive medications during the trial. For participants with CNS metastases, use of prednisone at a stable dose (or dose equivalent) of <= 20 mg/day is acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (111):
- Argentina (2):
  - Hospital Aleman, Caba
  - Centro Oncologico Riojano Integral (CORI), La Rioja
- Brazil (3):
  - CETUS Hospital Dia Oncologia, Uberaba, Minas Gerais
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
- China (5):
  - Beijing Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Shandong Cancer Hospital, Jinan
  - First Affiliated Hospital of Soochow University, Suzhou
  - Henan Cancer Hospital, Zhengzhou
- Organizacion Sanitas Internacional, Bogota, D.C., Colombia
- Clinica CIMCA, San José, Costa Rica
- Denmark (3):
  - Sjællands Universitetshospital, Næstved; Onkologisk Afdeling, Næstved
  - Odense Universitetshospital, Onkologisk Afdeling R, Odense C
  - Vejle Sygehus; Onkologisk Afdeling, Vejle
- Greece (6):
  - Anticancer Hospital Ag Savas; 1St Dept of Internal Medicine, Athens
  - Uoa Sotiria Hospital; Oncology, Athens
  - Agioi Anargyroi; 3Rd Dept. of Medical Oncology, Athens
  - Univ General Hosp Heraklion; Medical Oncology, Heraklion
  - University Hospital of Patras Medical Oncology, Pátrai
  - Diavalkaniko Hospital, Thessaloniki
- Oncomedica, Guatemala City, Guatemala
- Italy (16):
  - Ospedale Regionale Umberto Parini; S.C. Oncologia, Aosta, Aosta Valley
  - Ist. Ricovero e Cura a Carattere Scientifico-Centro Rif. Oncologico della Basilica, Rionero in Vulture (PZ), Basilicate
  - Campus Universitario S.Venuta; Centro Oncologico T.Campanella, Catanzaro, Calabria
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi; Unità Operativa Oncologia Medica, Bologna, Emilia-Romagna
  - Arcispedale Santa Maria Nuova; Medicina Nucleare, Reggio Emilia, Emilia-Romagna
  - Policlinico Umberto i di Roma; dip. Scienze Radiologiche, Oncologiche, Anatomopatologiche, Rome, Lazio
  - AZ. Ospedaliera San Giovanni - Addolorata, Rome, Lazio
  - Cliniche Gavazzeni S.p.A.; Dip. di Oncologia Pneumologica ed Urologica, Bergamo, Lombardy
  - ASST DEGLI SPEDALI CIVILI DI BRESCIA; Oncologia Medica, Brescia, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - Ospedale Oncologico A.Businco; Div. Oncologia Medica II, Cagliari, Sardinia
  - Ospedale Cannizzaro, Oncologia, Catania, Sicily
  - Ospedali Riuniti Di Ancona; Oncology, Ancona, The Marches
  - Azienda Ospedaliero-Universitaria Careggi; SOD Radioterapia, Florence, Tuscany
  - Azienda Ospedaliera Universitaria Pisana - Ospedale Cisanello; Dipartimento Cardio Toraco Vascolare, Pisa, Tuscany
  - ULSS2 Marca Trevigiana; UOC Oncologia Medica - Distretto di Treviso, Treviso, Veneto
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, R?ga
  - Riga East Clinical University Hospital Latvian Oncology Centre, Riga
- Lebanon (2):
  - Hotel Dieu de France; Oncology, Beirut
  - Bellevue Medical Center, El-Metn
- Malaysia (5):
  - University Malaya Medical Centre; Clinical Oncology Unit,, Kuala Lumpur, FED. Territory of Kuala Lumpur
  - Institute Kanser Negara (IKN), Putrajaya, FED. Territory of Kuala Lumpur
  - Hospital Pulau Pinang; Jabatan Respiratori, George Town, Pulau Pinang
  - Mount Miriam Cancer Hospital, Pulau Pinang, Pulau Pinang
  - Hospital Umum Sarawak; Oncology and Radiotherapy, Kuching, Sarawak
- Mexico (5):
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - Centro Oncologico Internacional, Mexico City, Mexico CITY (federal District)
  - Oaxaca Site Management Organization, Oaxaca City, Oaxaca
  - Oncologico Potosino, San Luis Potosí City, San Luis Potosí
  - Investigacion Clinica Merida, Mérida, Yucatán
- Morocco (3):
  - Clinique le Littoral, Casablanca
  - Centre Hospitalier Universitaire Hassan II, Fes
  - Institut National D'oncologie Sidi Med Benabdellah, Rabat
- Netherlands (6):
  - Meander Medisch Centrum, Amersfoort
  - Ziekenhuis Rijnstate, Arnhem
  - Amphia Ziekenhuis; Afdeling Longziekten, Breda
  - Tergooiziekenhuizen, loc. Hilversum, Hilversum
  - UMC Radboud Nijmegen, Nijmegen
  - Isala, Zwolle
- The Panama Clinic, Panama City, Panama
- Peru (2):
  - Instituto Regional de Enfermedades Neoplásicas del Sur; Centro de Inv. de Medicina Oncológica, Arequipa
  - Clinica Internacional, Sede San Borja; Unidad de Investigacion de Clínica Internacional, Lima
- Philippines (3):
  - University of Perpetual Help System DALTA Medical Center, Las Piñas
  - The Medical City Hospital; Cancer Research Room, Pasig
  - East Avenue Medical Center, Quezon City
- Poland (5):
  - Narodowy Instytut Onkologii Oddzial Gliwice; II Klinika Radioterapii i Chemioterapii, Gliwice
  - Samodzielny Publiczny Zespol Gruzlicy i Chorob Pluc w Olsztynie, Olsztyn
  - Mazowieckie Centrum Leczenia Chorob Pluc I Gruzlicy; Oddzial Iii, Otwock
  - Szpital Kliniczny; Przemienienia Panskiego;Uniwersytetu Medyczny im.; Karola Marcinkowskiego w Pozna, Poznan
  - Narod.Inst.Onkol. im. M.Sklodowskiej - Curie-Panst.Inst.Bad; Klinika Nowot.Pluca i Klatki Piers, Warsaw
- University Clinic Golnik, Golnik, Slovenia
- Spain (27):
  - Hospital Universitario Son Espases; Servicio de Oncologia, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Marques de Valdecilla; Servicio de Oncologia, Santander, Cantabria
  - Hospital Provincial de Castellon; Servicio de Oncologia, Castellon, Castellon
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Hospital de Donostia; Servicio de Oncologia Medica, Donostia / San Sebastian, Guipuzcoa
  - Complejo Hospitalario Universitario Insular?Materno Infantil; Servicio de Oncologia, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Universitario Puerta de Hierro; Servicio de Oncologia, Majadahonda, Madrid
  - Hospital Quiron de Madrid; Servicio de Oncologia, Pozuelo de Alarcón, Madrid
  - Hospital Infanta Sofia; Servico de Oncologia, San Sebastián de los Reyes, Madrid
  - Complejo Hospitalario de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Hospital Univ. Central de Asturias; Servicio de Oncologia, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias;servicio de Oncologia, San Cristóbal de La Laguna, Tenerife
  - Hospital General Univ. de Alicante; Servicio de Oncologia, Alicante
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Oncologia, Barcelona
  - Hospital Universitari de Girona Dr Josep Trueta; Departamento de Oncologia Medica, Girona
  - Hospital Universitario Virgen de las Nieves; Servicio de Oncologia, Granada
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico; Servicio de Oncologia, Jaén
  - Hospital Lucus Augusti; Servicio de Oncologia, Lugo
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
  - Hospital General Universitario de Valencia; Servicio de oncologia, Valencia
  - Hospital Universitario la Fe; Servicio de Oncologia, Valencia
  - Hospital Clinico Universitario Lozano Blesa; Servicio de Oncologia, Zaragoza
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Lungmedicinkliniken, Gothenburg
  - Karolinska Universitetssjukhuset, Solna; Kliniska prövningsenheten Z:4:01, Stockholm
  - Uppsala University Hospital; Department of Oncology, Uppsala
- Tawam Hospital, Al Ain City, United Arab Emirates
- United Kingdom (7):
  - Royal United Hospital, Bath
  - Birmingham Heartlands Hospital ; Department of Respiratory Medicine (Rm 30), Birmingham
  - Castle Hill Hospital; The Queen's Centre for Oncology & Haematology, Hull
  - Forth Valley Royal Hospital ; Oncology Department, Larbert
  - Chelsea & Westminster Hospital, London
  - Mount Vernon Cancer Centre, Northwood
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Ardizzoni A, Azevedo S, Rubio-Viqueira B, Rodriguez-Abreu D, Alatorre-Alexander J, Smit HJM, Yu J, Syrigos K, Hoglander E, Kaul M, Tolson J, Hu Y, Vollan HK, Newsom-Davis T. Final results from TAIL: updated long-term efficacy of atezolizumab in a diverse population of patients with previously treated advanced non-small cell lung cancer. J Immunother Cancer. 2022 Nov;10(11):e005581. doi: 10.1136/jitc-2022-005581. PMID 36450379
- [Derived] Ardizzoni A, Azevedo S, Rubio-Viqueira B, Rodriguez-Abreu D, Alatorre-Alexander J, Smit HJM, Yu J, Syrigos K, Trunzer K, Patel H, Tolson J, Cardona A, Perez-Moreno PD, Newsom-Davis T. Primary results from TAIL: a global single-arm safety study of atezolizumab monotherapy in a diverse population of patients with previously treated advanced non-small cell lung cancer. J Immunother Cancer. 2021 Mar;9(3):e001865. doi: 10.1136/jitc-2020-001865. PMID 33737339

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 111 sites across 24 countries.
Pre-assignment Details: Four enrolled participants died without receiving study treatment.
Groups:
- Atezolizumab: Participants with Stage IIIb or State IV NSCLC who had progressed after standard systemic chemotherapy received atezolizumab until Investigator-assessed loss of clinical benefit, unacceptable toxicity, investigator or participant's decision to withdraw from therapy, or death (whichever occurred first).
Period: Overall Study
Arm/Group | Atezolizumab
Started | 615
Completed | 13
Not Completed | 602
Not completed — Death | 470
Not completed — Lost to Follow-up | 18
Not completed — Physician Decision | 2
Not completed — Study Terminated By Sponsor | 79
Not completed — Withdrawal by Subject | 33

BASELINE CHARACTERISTICS:
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245
  Male | 370
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 93
  Not Hispanic or Latino | 509
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 44
  Asian | 76
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 483
  More than one race | 5
  Unknown or Not Reported | 2
Region [Count of Participants; unit: Participants]
  EMEA (Europe, the Middle East, and Africa) | 455
  Asia | 70
  LATAM (Latin America) | 90
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status is graded from 0-5 with a lower number representing no or limited impact on daily living activities and a higher number represents greater impact on daily living activities.
  Participants
    ECOG performance status 0 (fully active) | 193
    ECOG performance status 1 (restricted in physically strenuous activity) | 361
    ECOG performance status 2 (ambulatory and capable of selfcare; unable to carry out work activities) | 61
Smoking Status [Count of Participants; unit: Participants]
  Never | 127
  Current | 115
  Previous | 373
eGFR (mL/min/1.73 m^2) at baseline [Count of Participants; unit: Participants]
  15-<30 | 2
  30-<60 | 77
  60-<90 | 251
  >=90 | 283
  Missing | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unitended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a pharmaceutical product whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as a AEs.
Time Frame: Baseline up to 4 years
Population: The safety population was based on all participants who received any dose of atezolizumab during the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Participants | 564

2. Secondary Outcome: Percentage of Participants Alive 2 Years After Initiation of Treatment
Description: The overall survival (OS) rate at 2 years, was defined as the percentage of participants remaining alive 2 years after initiation of study treatment.
Time Frame: Baseline up to Year 2
Population: The safety population was based on all participants who received any dose of atezolizumab during the study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Percentage of Participants | 26.7

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (in months) from initiation of study treatment to death from any cause.
Time Frame: Baseline up to death (up to 4 years)
Population: The safety population was based on all participants who received any dose of atezolizumab during the study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Months | 11.2 [8.9 to 12.7]

4. Secondary Outcome: Progression-Free Survival (PFS) as Evaluated By the Investigator in Accordance With Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 (v.1.1)
Description: PFS was defined as the time (in months) from initiation of study treatment to the first documented disease progression or death from any cause, whichever occurred first. PFS was evaluated by the investigator according to RECIST v1.1.
Time Frame: Baseline up to disease progression or death whichever occurs first (up to 4 years)
Population: The safety population was based on all participants who received any dose of atezolizumab during the study treatment. This was a single-arm study. The study population was participants with Stage IIIB or Stage IV NSCLC. The primary objective of this study was to understand the safety in this participant population (without distinction of Stage IIIB and IV) and it was not planned to analyze them separately as per the protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Months | 2.7 [2.3 to 2.8]

5. Secondary Outcome: EuroQol 5-Dimension 5-Level (EQ-5D-5L) Questionnaire - Mobility Item
Description: The EQ-5D-5L was a self-reported health status questionnaire that consisted of six questions used to calculate a health utility score for use in health economic analysis. The EQ-5D-5L has two components: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, as well as a Visual Analogue Scale (VAS) that measures health state. Each item was rated from 1 (no problems) to 5 (extreme problems). Categories with non-zero values are reported here. Number of participants who rated the mobility item ranging from 1-5 are reported. Participants who had a invalid response were presented under the category 'Invalid Response'.
Time Frame: Day 1 of first 2 cycles (21-day cycle), then every 6 weeks for 54 weeks; thereafter every 3 weeks or 6 weeks until disease progression or until treatment discontinuation (up to 4 years)
Population: The safety population was based on all participants who received any dose of atezolizumab during the study treatment. Number analyzed are unique number of participants out of all the assessed participants who were evaluable at specified timepoint. Different participants may have contributed data for each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Participants
  Baseline: No Problem: number analyzed (Participants) | 597
  Baseline: No Problem | 328
  Baseline: Slight Problem: number analyzed (Participants) | 597
  Baseline: Slight Problem | 146
  Baseline: Moderate Problems: number analyzed (Participants) | 597
  Baseline: Moderate Problems | 97
  Baseline: Severe Problems: number analyzed (Participants) | 597
  Baseline: Severe Problems | 24
  Baseline: Extreme Problems: number analyzed (Participants) | 597
  Baseline: Extreme Problems | 1
  Baseline: Invalid Response: number analyzed (Participants) | 597
  Baseline: Invalid Response | 1
  Cycle 2 Day 1: No Problem: number analyzed (Participants) | 534
  Cycle 2 Day 1: No Problem | 274
  Cycle 2 Day 1: Slight Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Slight Problems | 145
  Cycle 2 Day 1: Moderate Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Moderate Problems | 84
  Cycle 2 Day 1: Severe Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Severe Problems | 26
  Cycle 2 Day 1: Extreme Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Extreme Problems | 4
  Cycle 2 Day 1: Invalid Response: number analyzed (Participants) | 534
  Cycle 2 Day 1: Invalid Response | 1
  Tumor Assessment Week 006: No Problem: number analyzed (Participants) | 438
  Tumor Assessment Week 006: No Problem | 229
  Tumor Assessment Week 006: Slight Problems: number analyzed (Participants) | 438
  Tumor Assessment Week 006: Slight Problems | 121
  Tumor Assessment Week 006: Moderate Problems: number analyzed (Participants) | 438
  Tumor Assessment Week 006: Moderate Problems | 69
  Tumor Assessment Week 006: Severe Problems: number analyzed (Participants) | 438
  Tumor Assessment Week 006: Severe Problems | 16
  Tumor Assessment Week 006: Extreme Problems: number analyzed (Participants) | 438
  Tumor Assessment Week 006: Extreme Problems | 3
  Tumor Assessment Week 012: No Problem: number analyzed (Participants) | 323
  Tumor Assessment Week 012: No Problem | 183
  Tumor Assessment Week 012: Slight Problems: number analyzed (Participants) | 323
  Tumor Assessment Week 012: Slight Problems | 75
  Tumor Assessment Week 012: Moderate Problems: number analyzed (Participants) | 323
  Tumor Assessment Week 012: Moderate Problems | 48
  Tumor Assessment Week 012: Severe Problems: number analyzed (Participants) | 323
  Tumor Assessment Week 012: Severe Problems | 10
  Tumor Assessment Week 012: Extreme Problems: number analyzed (Participants) | 323
  Tumor Assessment Week 012: Extreme Problems | 5
  Tumor Assessment Week 012: Invalid Response: number analyzed (Participants) | 323
  Tumor Assessment Week 012: Invalid Response | 2
  Tumor Assessment Week 018: No Problem: number analyzed (Participants) | 260
  Tumor Assessment Week 018: No Problem | 153
  Tumor Assessment Week 018: Slight Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Slight Problems | 66
  Tumor Assessment Week 018: Moderate Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Moderate Problems | 27
  Tumor Assessment Week 018: Severe Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Severe Problems | 11
  Tumor Assessment Week 018: Extreme Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Extreme Problems | 3
  Tumor Assessment Week 024: No Problem: number analyzed (Participants) | 220
  Tumor Assessment Week 024: No Problem | 131
  Tumor Assessment Week 024: Slight Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Slight Problems | 56
  Tumor Assessment Week 024: Moderate Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Moderate Problems | 22
  Tumor Assessment Week 024: Severe Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Severe Problems | 4
  Tumor Assessment Week 024: Extreme Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Extreme Problems | 4
  Tumor Assessment Week 024: Invalid Response: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Invalid Response | 3
  Tumor Assessment Week 030: No Problem: number analyzed (Participants) | 184
  Tumor Assessment Week 030: No Problem | 124
  Tumor Assessment Week 030: Slight Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Slight Problems | 41
  Tumor Assessment Week 030: Moderate Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Moderate Problems | 14
  Tumor Assessment Week 030: Severe Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Severe Problems | 4
  Tumor Assessment Week 030: Extreme Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Extreme Problems | 1
  Tumor Assessment Week 036: No Problem: number analyzed (Participants) | 162
  Tumor Assessment Week 036: No Problem | 110
  Tumor Assessment Week 036: Slight Problems: number analyzed (Participants) | 162
  Tumor Assessment Week 036: Slight Problems | 31
  Tumor Assessment Week 036: Moderate Problems: number analyzed (Participants) | 162
  Tumor Assessment Week 036: Moderate Problems | 20
  Tumor Assessment Week 036: Severe Problems: number analyzed (Participants) | 162
  Tumor Assessment Week 036: Severe Problems | 1
  Tumor Assessment Week 042: No Problem: number analyzed (Participants) | 145
  Tumor Assessment Week 042: No Problem | 88
  Tumor Assessment Week 042: Slight Problems: number analyzed (Participants) | 145
  Tumor Assessment Week 042: Slight Problems | 39
  Tumor Assessment Week 042: Moderate Problems: number analyzed (Participants) | 145
  Tumor Assessment Week 042: Moderate Problems | 14
  Tumor Assessment Week 042: Severe Problems: number analyzed (Participants) | 145
  Tumor Assessment Week 042: Severe Problems | 4
  Tumor Assessment Week 048: No Problem: number analyzed (Participants) | 127
  Tumor Assessment Week 048: No Problem | 75
  Tumor Assessment Week 048: Slight Problems: number analyzed (Participants) | 127
  Tumor Assessment Week 048: Slight Problems | 32
  Tumor Assessment Week 048: Moderate Problems: number analyzed (Participants) | 127
  Tumor Assessment Week 048: Moderate Problems | 16
  Tumor Assessment Week 048: Severe Problems: number analyzed (Participants) | 127
  Tumor Assessment Week 048: Severe Problems | 3
  Tumor Assessment Week 048: Extreme Problems: number analyzed (Participants) | 127
  Tumor Assessment Week 048: Extreme Problems | 1
  Tumor Assessment Week 054: No Problem: number analyzed (Participants) | 23
  Tumor Assessment Week 054: No Problem | 11
  Tumor Assessment Week 054: Slight Problems: number analyzed (Participants) | 23
  Tumor Assessment Week 054: Slight Problems | 6
  Tumor Assessment Week 054: Moderate Problems: number analyzed (Participants) | 23
  Tumor Assessment Week 054: Moderate Problems | 5
  Tumor Assessment Week 054: Severe Problems: number analyzed (Participants) | 23
  Tumor Assessment Week 054: Severe Problems | 1
  Tumor Assessment Week 057: No Problem: number analyzed (Participants) | 97
  Tumor Assessment Week 057: No Problem | 64
  Tumor Assessment Week 057: Slight Problems: number analyzed (Participants) | 97
  Tumor Assessment Week 057: Slight Problems | 20
  Tumor Assessment Week 057: Moderate Problems: number analyzed (Participants) | 97
  Tumor Assessment Week 057: Moderate Problems | 8
  Tumor Assessment Week 057: Severe Problems: number analyzed (Participants) | 97
  Tumor Assessment Week 057: Severe Problems | 3
  Tumor Assessment Week 057: Extreme Problems: number analyzed (Participants) | 97
  Tumor Assessment Week 057: Extreme Problems | 2
  Tumor Assessment Week 060: No Problem: number analyzed (Participants) | 17
  Tumor Assessment Week 060: No Problem | 10
  Tumor Assessment Week 060: Slight Problems: number analyzed (Participants) | 17
  Tumor Assessment Week 060: Slight Problems | 3
  Tumor Assessment Week 060: Moderate Problems: number analyzed (Participants) | 17
  Tumor Assessment Week 060: Moderate Problems | 3
  Tumor Assessment Week 060: Extreme Problems: number analyzed (Participants) | 17
  Tumor Assessment Week 060: Extreme Problems | 1
  Tumor Assessment Week 066: No Problem: number analyzed (Participants) | 88
  Tumor Assessment Week 066: No Problem | 56
  Tumor Assessment Week 066: Slight Problems: number analyzed (Participants) | 88
  Tumor Assessment Week 066: Slight Problems | 20
  Tumor Assessment Week 066: Moderate Problems: number analyzed (Participants) | 88
  Tumor Assessment Week 066: Moderate Problems | 9
  Tumor Assessment Week 066: Severe Problems: number analyzed (Participants) | 88
  Tumor Assessment Week 066: Severe Problems | 2
  Tumor Assessment Week 066: Extreme Problems: number analyzed (Participants) | 88
  Tumor Assessment Week 066: Extreme Problems | 1
  Tumor Assessment Week 072: No Problem: number analyzed (Participants) | 13
  Tumor Assessment Week 072: No Problem | 7
  Tumor Assessment Week 072: Slight Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 072: Slight Problems | 4
  Tumor Assessment Week 072: Moderate Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 072: Moderate Problems | 2
  Tumor Assessment Week 075: No Problem: number analyzed (Participants) | 73
  Tumor Assessment Week 075: No Problem | 45
  Tumor Assessment Week 075: Slight Problems: number analyzed (Participants) | 73
  Tumor Assessment Week 075: Slight Problems | 20
  Tumor Assessment Week 075: Moderate Problems: number analyzed (Participants) | 73
  Tumor Assessment Week 075: Moderate Problems | 7
  Tumor Assessment Week 075: Severe Problems: number analyzed (Participants) | 73
  Tumor Assessment Week 075: Severe Problems | 1
  Tumor Assessment Week 078: No Problem: number analyzed (Participants) | 10
  Tumor Assessment Week 078: No Problem | 6
  Tumor Assessment Week 078: Slight Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 078: Slight Problems | 3
  Tumor Assessment Week 078: Severe Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 078: Severe Problems | 1
  Tumor Assessment Week 084: No Problem: number analyzed (Participants) | 67
  Tumor Assessment Week 084: No Problem | 47
  Tumor Assessment Week 084: Slight Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Slight Problems | 12
  Tumor Assessment Week 084: Moderate Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Moderate Problems | 6
  Tumor Assessment Week 084: Severe Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Severe Problems | 2
  Tumor Assessment Week 090: No Problem: number analyzed (Participants) | 10
  Tumor Assessment Week 090: No Problem | 7
  Tumor Assessment Week 090: Slight Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 090: Slight Problems | 2
  Tumor Assessment Week 090: Moderate Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 090: Moderate Problems | 1
  Tumor Assessment Week 093: No Problem: number analyzed (Participants) | 53
  Tumor Assessment Week 093: No Problem | 34
  Tumor Assessment Week 093: Slight Problems: number analyzed (Participants) | 53
  Tumor Assessment Week 093: Slight Problems | 16
  Tumor Assessment Week 093: Moderate Problems: number analyzed (Participants) | 53
  Tumor Assessment Week 093: Moderate Problems | 2
  Tumor Assessment Week 093: Extreme Problems: number analyzed (Participants) | 53
  Tumor Assessment Week 093: Extreme Problems | 1
  Tumor Assessment Week 096: No Problem: number analyzed (Participants) | 7
  Tumor Assessment Week 096: No Problem | 4
  Tumor Assessment Week 096: Slight Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 096: Slight Problems | 2
  Tumor Assessment Week 096: Severe Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 096: Severe Problems | 1
  Tumor Assessment Week 102: No Problem: number analyzed (Participants) | 55
  Tumor Assessment Week 102: No Problem | 33
  Tumor Assessment Week 102: Slight Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Slight Problems | 16
  Tumor Assessment Week 102: Moderate Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Moderate Problems | 4
  Tumor Assessment Week 102: Severe Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Severe Problems | 1
  Tumor Assessment Week 102: Extreme Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Extreme Problems | 1
  Tumor Assessment Week 108: No Problem: number analyzed (Participants) | 7
  Tumor Assessment Week 108: No Problem | 3
  Tumor Assessment Week 108: Slight Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 108: Slight Problems | 3
  Tumor Assessment Week 108: Moderate Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 108: Moderate Problems | 1
  Tumor Assessment Week 111: No Problem: number analyzed (Participants) | 41
  Tumor Assessment Week 111: No Problem | 25
  Tumor Assessment Week 111: Slight Problems: number analyzed (Participants) | 41
  Tumor Assessment Week 111: Slight Problems | 13
  Tumor Assessment Week 111: Moderate Problems: number analyzed (Participants) | 41
  Tumor Assessment Week 111: Moderate Problems | 2
  Tumor Assessment Week 111: Severe Problems: number analyzed (Participants) | 41
  Tumor Assessment Week 111: Severe Problems | 1
  Tumor Assessment Week 114: Slight Problems: number analyzed (Participants) | 2
  Tumor Assessment Week 114: Slight Problems | 1
  Tumor Assessment Week 114: Moderate Problems: number analyzed (Participants) | 2
  Tumor Assessment Week 114: Moderate Problems | 1
  Tumor Assessment Week 120: No Problem: number analyzed (Participants) | 38
  Tumor Assessment Week 120: No Problem | 22
  Tumor Assessment Week 120: Slight Problems: number analyzed (Participants) | 38
  Tumor Assessment Week 120: Slight Problems | 14
  Tumor Assessment Week 120: Moderate Problems: number analyzed (Participants) | 38
  Tumor Assessment Week 120: Moderate Problems | 1
  Tumor Assessment Week 120: Extreme Problems: number analyzed (Participants) | 38
  Tumor Assessment Week 120: Extreme Problems | 1
  Tumor Assessment Week 126: No Problem: number analyzed (Participants) | 4
  Tumor Assessment Week 126: No Problem | 1
  Tumor Assessment Week 126: Slight Problems: number analyzed (Participants) | 4
  Tumor Assessment Week 126: Slight Problems | 3
  Tumor Assessment Week 129: No Problem: number analyzed (Participants) | 32
  Tumor Assessment Week 129: No Problem | 19
  Tumor Assessment Week 129: Slight Problems: number analyzed (Participants) | 32
  Tumor Assessment Week 129: Slight Problems | 11
  Tumor Assessment Week 129: Moderate Problems: number analyzed (Participants) | 32
  Tumor Assessment Week 129: Moderate Problems | 1
  Tumor Assessment Week 129: Severe Problems: number analyzed (Participants) | 32
  Tumor Assessment Week 129: Severe Problems | 1
  Tumor Assessment Week 132: No Problem: number analyzed (Participants) | 2
  Tumor Assessment Week 132: No Problem | 1
  Tumor Assessment Week 132: Slight Problems: number analyzed (Participants) | 2
  Tumor Assessment Week 132: Slight Problems | 1
  Tumor Assessment Week 138: No Problem: number analyzed (Participants) | 28
  Tumor Assessment Week 138: No Problem | 17
  Tumor Assessment Week 138: Slight Problems: number analyzed (Participants) | 28
  Tumor Assessment Week 138: Slight Problems | 10
  Tumor Assessment Week 138: Extreme Problems: number analyzed (Participants) | 28
  Tumor Assessment Week 138: Extreme Problems | 1
  Tumor Assessment Week 144: No Problem: number analyzed (Participants) | 1
  Tumor Assessment Week 144: No Problem | 1
  Tumor Assessment Week 147: No Problem: number analyzed (Participants) | 21
  Tumor Assessment Week 147: No Problem | 14
  Tumor Assessment Week 147: Slight Problems: number analyzed (Participants) | 21
  Tumor Assessment Week 147: Slight Problems | 6
  Tumor Assessment Week 147: Severe Problems: number analyzed (Participants) | 21
  Tumor Assessment Week 147: Severe Problems | 1
  Tumor Assessment Week 156: No Problem: number analyzed (Participants) | 15
  Tumor Assessment Week 156: No Problem | 8
  Tumor Assessment Week 156: Slight Problems: number analyzed (Participants) | 15
  Tumor Assessment Week 156: Slight Problems | 5
  Tumor Assessment Week 156: Moderate Problems: number analyzed (Participants) | 15
  Tumor Assessment Week 156: Moderate Problems | 1
  Tumor Assessment Week 156: Severe Problems: number analyzed (Participants) | 15
  Tumor Assessment Week 156: Severe Problems | 1
  Tumor Assessment Week 165: No Problem: number analyzed (Participants) | 13
  Tumor Assessment Week 165: No Problem | 3
  Tumor Assessment Week 165: Slight Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Slight Problems | 8
  Tumor Assessment Week 165: Severe Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Severe Problems | 1
  Tumor Assessment Week 165: Invalid Response: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Invalid Response | 1
  Tumor Assessment Week 174: No Problem: number analyzed (Participants) | 10
  Tumor Assessment Week 174: No Problem | 6
  Tumor Assessment Week 174: Slight Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 174: Slight Problems | 4
  Tumor Assessment Week 183: Slight Problems: number analyzed (Participants) | 3
  Tumor Assessment Week 183: Slight Problems | 3

6. Secondary Outcome: EQ-5D-5L Questionnaire - Self-Care Item
Description: The EQ-5D-5L was a self-reported health status questionnaire that consisted of six questions used to calculate a health utility score for use in health economic analysis. The EQ-5D-5L has two components: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, as well as a VAS that measures health state. Each item was rated from 1 (no problems) to 5 (extreme problems). Categories with non-zero values are reported here. Number of participants who rated the self-care item ranging from 1-5 are reported. Participants who had a invalid response were presented under the category 'Invalid Response'.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Participants
  Baseline: No Problem: number analyzed (Participants) | 598
  Baseline: No Problem | 475
  Baseline: Slight Problem: number analyzed (Participants) | 598
  Baseline: Slight Problem | 66
  Baseline: Moderate Problems: number analyzed (Participants) | 598
  Baseline: Moderate Problems | 44
  Baseline: Severe Problems: number analyzed (Participants) | 598
  Baseline: Severe Problems | 8
  Baseline: Extreme Problems: number analyzed (Participants) | 598
  Baseline: Extreme Problems | 4
  Baseline: Invalid Response: number analyzed (Participants) | 598
  Baseline: Invalid Response | 1
  Cycle 2 Day 1: No Problem: number analyzed (Participants) | 534
  Cycle 2 Day 1: No Problem | 402
  Cycle 2 Day 1: Slight Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Slight Problems | 79
  Cycle 2 Day 1: Moderate: number analyzed (Participants) | 534
  Cycle 2 Day 1: Moderate | 37
  Cycle 2 Day 1: Severe Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Severe Problems | 10
  Cycle 2 Day 1: Extreme Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Extreme Problems | 5
  Cycle 2 Day 1: Invalid Response: number analyzed (Participants) | 534
  Cycle 2 Day 1: Invalid Response | 1
  Tumor Assessment Week 006: No Problem: number analyzed (Participants) | 438
  Tumor Assessment Week 006: No Problem | 327
  Tumor Assessment Week 006: Slight Problems: number analyzed (Participants) | 438
  Tumor Assessment Week 006: Slight Problems | 67
  Tumor Assessment Week 006: Moderate Problems: number analyzed (Participants) | 438
  Tumor Assessment Week 006: Moderate Problems | 33
  Tumor Assessment Week 006: Severe Problems: number analyzed (Participants) | 438
  Tumor Assessment Week 006: Severe Problems | 6
  Tumor Assessment Week 006: Extreme Problems: number analyzed (Participants) | 438
  Tumor Assessment Week 006: Extreme Problems | 5
  Tumor Assessment Week 012: No Problem: number analyzed (Participants) | 322
  Tumor Assessment Week 012: No Problem | 245
  Tumor Assessment Week 012: Slight Problems: number analyzed (Participants) | 322
  Tumor Assessment Week 012: Slight Problems | 47
  Tumor Assessment Week 012: Moderate Problems: number analyzed (Participants) | 322
  Tumor Assessment Week 012: Moderate Problems | 20
  Tumor Assessment Week 012: Severe Problems: number analyzed (Participants) | 322
  Tumor Assessment Week 012: Severe Problems | 5
  Tumor Assessment Week 012: Extreme Problems: number analyzed (Participants) | 322
  Tumor Assessment Week 012: Extreme Problems | 5
  Tumor Assessment Week 018: No Problem: number analyzed (Participants) | 260
  Tumor Assessment Week 018: No Problem | 205
  Tumor Assessment Week 018: Slight Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Slight Problems | 35
  Tumor Assessment Week 018: Moderate Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Moderate Problems | 16
  Tumor Assessment Week 018: Severe Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Severe Problems | 2
  Tumor Assessment Week 018: Extreme Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Extreme Problems | 2
  Tumor Assessment Week 024: No Problem: number analyzed (Participants) | 220
  Tumor Assessment Week 024: No Problem | 174
  Tumor Assessment Week 024: Slight Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Slight Problems | 35
  Tumor Assessment Week 024: Moderate Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Moderate Problems | 5
  Tumor Assessment Week 024: Severe Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Severe Problems | 1
  Tumor Assessment Week 024: Extreme Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Extreme Problems | 2
  Tumor Assessment Week 024: Invalid Response: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Invalid Response | 3
  Tumor Assessment Week 030: No Problem: number analyzed (Participants) | 184
  Tumor Assessment Week 030: No Problem | 150
  Tumor Assessment Week 030: Slight Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Slight Problems | 26
  Tumor Assessment Week 030: Moderate Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Moderate Problems | 7
  Tumor Assessment Week 030: Extreme Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Extreme Problems | 1
  Tumor Assessment Week 036: No Problem: number analyzed (Participants) | 162
  Tumor Assessment Week 036: No Problem | 129
  Tumor Assessment Week 036: Slight Problems: number analyzed (Participants) | 162
  Tumor Assessment Week 036: Slight Problems | 24
  Tumor Assessment Week 036: Moderate Problems: number analyzed (Participants) | 162
  Tumor Assessment Week 036: Moderate Problems | 9
  Tumor Assessment Week 042: No Problem: number analyzed (Participants) | 145
  Tumor Assessment Week 042: No Problem | 113
  Tumor Assessment Week 042: Slight Problems: number analyzed (Participants) | 145
  Tumor Assessment Week 042: Slight Problems | 23
  Tumor Assessment Week 042: Moderate Problems: number analyzed (Participants) | 145
  Tumor Assessment Week 042: Moderate Problems | 9
  Tumor Assessment Week 048: No Problem: number analyzed (Participants) | 127
  Tumor Assessment Week 048: No Problem | 99
  Tumor Assessment Week 048: Slight Problems: number analyzed (Participants) | 127
  Tumor Assessment Week 048: Slight Problems | 18
  Tumor Assessment Week 048: Moderate Problems: number analyzed (Participants) | 127
  Tumor Assessment Week 048: Moderate Problems | 8
  Tumor Assessment Week 048: Severe Problems: number analyzed (Participants) | 127
  Tumor Assessment Week 048: Severe Problems | 2
  Tumor Assessment Week 054: No Problem: number analyzed (Participants) | 23
  Tumor Assessment Week 054: No Problem | 15
  Tumor Assessment Week 054: Slight Problems: number analyzed (Participants) | 23
  Tumor Assessment Week 054: Slight Problems | 5
  Tumor Assessment Week 054: Moderate Problems: number analyzed (Participants) | 23
  Tumor Assessment Week 054: Moderate Problems | 3
  Tumor Assessment Week 057: No Problem: number analyzed (Participants) | 96
  Tumor Assessment Week 057: No Problem | 78
  Tumor Assessment Week 057: Slight Problems: number analyzed (Participants) | 96
  Tumor Assessment Week 057: Slight Problems | 12
  Tumor Assessment Week 057: Moderate Problems: number analyzed (Participants) | 96
  Tumor Assessment Week 057: Moderate Problems | 5
  Tumor Assessment Week 057: Extreme Problems: number analyzed (Participants) | 96
  Tumor Assessment Week 057: Extreme Problems | 1
  Tumor Assessment Week 060: No Problem: number analyzed (Participants) | 17
  Tumor Assessment Week 060: No Problem | 12
  Tumor Assessment Week 060: Slight Problems: number analyzed (Participants) | 17
  Tumor Assessment Week 060: Slight Problems | 4
  Tumor Assessment Week 060: Moderate Problems: number analyzed (Participants) | 17
  Tumor Assessment Week 060: Moderate Problems | 1
  Tumor Assessment Week 066: No Problem: number analyzed (Participants) | 88
  Tumor Assessment Week 066: No Problem | 69
  Tumor Assessment Week 066: Slight Problems: number analyzed (Participants) | 88
  Tumor Assessment Week 066: Slight Problems | 14
  Tumor Assessment Week 066: Moderate Problems: number analyzed (Participants) | 88
  Tumor Assessment Week 066: Moderate Problems | 5
  Tumor Assessment Week 072: No Problem: number analyzed (Participants) | 13
  Tumor Assessment Week 072: No Problem | 10
  Tumor Assessment Week 072: Slight Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 072: Slight Problems | 3
  Tumor Assessment Week 075: No Problem: number analyzed (Participants) | 73
  Tumor Assessment Week 075: No Problem | 57
  Tumor Assessment Week 075: Slight Problems: number analyzed (Participants) | 73
  Tumor Assessment Week 075: Slight Problems | 14
  Tumor Assessment Week 075: Moderate Problems: number analyzed (Participants) | 73
  Tumor Assessment Week 075: Moderate Problems | 1
  Tumor Assessment Week 075: Extreme Problems: number analyzed (Participants) | 73
  Tumor Assessment Week 075: Extreme Problems | 1
  Tumor Assessment Week 078: No Problem: number analyzed (Participants) | 10
  Tumor Assessment Week 078: No Problem | 7
  Tumor Assessment Week 078: Slight Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 078: Slight Problems | 2
  Tumor Assessment Week 078: Severe Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 078: Severe Problems | 1
  Tumor Assessment Week 084: No Problem: number analyzed (Participants) | 67
  Tumor Assessment Week 084: No Problem | 51
  Tumor Assessment Week 084: Slight Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Slight Problems | 12
  Tumor Assessment Week 084: Moderate Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Moderate Problems | 3
  Tumor Assessment Week 084: Severe Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Severe Problems | 1
  Tumor Assessment Week 090: No Problem: number analyzed (Participants) | 10
  Tumor Assessment Week 090: No Problem | 6
  Tumor Assessment Week 090: Slight Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 090: Slight Problems | 3
  Tumor Assessment Week 090: Severe Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 090: Severe Problems | 1
  Tumor Assessment Week 093: No Problem: number analyzed (Participants) | 53
  Tumor Assessment Week 093: No Problem | 44
  Tumor Assessment Week 093: Slight Problems: number analyzed (Participants) | 53
  Tumor Assessment Week 093: Slight Problems | 7
  Tumor Assessment Week 093: Severe Problems: number analyzed (Participants) | 53
  Tumor Assessment Week 093: Severe Problems | 1
  Tumor Assessment Week 093: Extreme Problems: number analyzed (Participants) | 53
  Tumor Assessment Week 093: Extreme Problems | 1
  Tumor Assessment Week 096: No Problem: number analyzed (Participants) | 7
  Tumor Assessment Week 096: No Problem | 4
  Tumor Assessment Week 096: Slight Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 096: Slight Problems | 2
  Tumor Assessment Week 096: Severe Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 096: Severe Problems | 1
  Tumor Assessment Week 102: No Problem: number analyzed (Participants) | 55
  Tumor Assessment Week 102: No Problem | 45
  Tumor Assessment Week 102: Slight Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Slight Problems | 7
  Tumor Assessment Week 102: Moderate Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Moderate Problems | 1
  Tumor Assessment Week 102: Severe Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Severe Problems | 1
  Tumor Assessment Week 102: Extreme Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Extreme Problems | 1
  Tumor Assessment Week 108: No Problem: number analyzed (Participants) | 7
  Tumor Assessment Week 108: No Problem | 3
  Tumor Assessment Week 108: Slight Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 108: Slight Problems | 4
  Tumor Assessment Week 111: No Problem: number analyzed (Participants) | 41
  Tumor Assessment Week 111: No Problem | 33
  Tumor Assessment Week 111: Slight Problems: number analyzed (Participants) | 41
  Tumor Assessment Week 111: Slight Problems | 7
  Tumor Assessment Week 111: Extreme Problems: number analyzed (Participants) | 41
  Tumor Assessment Week 111: Extreme Problems | 1
  Tumor Assessment Week 114: Slight Problems: number analyzed (Participants) | 2
  Tumor Assessment Week 114: Slight Problems | 1
  Tumor Assessment Week 114: Moderate Problems: number analyzed (Participants) | 2
  Tumor Assessment Week 114: Moderate Problems | 1
  Tumor Assessment Week 120: No Problem: number analyzed (Participants) | 38
  Tumor Assessment Week 120: No Problem | 30
  Tumor Assessment Week 120: Slight Problems: number analyzed (Participants) | 38
  Tumor Assessment Week 120: Slight Problems | 7
  Tumor Assessment Week 120: Moderate Problems: number analyzed (Participants) | 38
  Tumor Assessment Week 120: Moderate Problems | 1
  Tumor Assessment Week 126: No Problem: number analyzed (Participants) | 4
  Tumor Assessment Week 126: No Problem | 1
  Tumor Assessment Week 126: Slight Problems: number analyzed (Participants) | 4
  Tumor Assessment Week 126: Slight Problems | 3
  Tumor Assessment Week 129: No Problem: number analyzed (Participants) | 32
  Tumor Assessment Week 129: No Problem | 26
  Tumor Assessment Week 129: Slight Problems: number analyzed (Participants) | 32
  Tumor Assessment Week 129: Slight Problems | 5
  Tumor Assessment Week 129: Extreme Problems: number analyzed (Participants) | 32
  Tumor Assessment Week 129: Extreme Problems | 1
  Tumor Assessment Week 132: No Problem: number analyzed (Participants) | 2
  Tumor Assessment Week 132: No Problem | 1
  Tumor Assessment Week 132: Slight Problems: number analyzed (Participants) | 2
  Tumor Assessment Week 132: Slight Problems | 1
  Tumor Assessment Week 138: No Problem: number analyzed (Participants) | 28
  Tumor Assessment Week 138: No Problem | 23
  Tumor Assessment Week 138: Slight Problems: number analyzed (Participants) | 28
  Tumor Assessment Week 138: Slight Problems | 5
  Tumor Assessment Week 144: No Problem: number analyzed (Participants) | 1
  Tumor Assessment Week 144: No Problem | 1
  Tumor Assessment Week 147: No Problem: number analyzed (Participants) | 21
  Tumor Assessment Week 147: No Problem | 19
  Tumor Assessment Week 147: Slight Problems: number analyzed (Participants) | 21
  Tumor Assessment Week 147: Slight Problems | 2
  Tumor Assessment Week 156: No Problem: number analyzed (Participants) | 15
  Tumor Assessment Week 156: No Problem | 11
  Tumor Assessment Week 156: Slight Problems: number analyzed (Participants) | 15
  Tumor Assessment Week 156: Slight Problems | 4
  Tumor Assessment Week 165: No Problem: number analyzed (Participants) | 13
  Tumor Assessment Week 165: No Problem | 10
  Tumor Assessment Week 165: Slight Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Slight Problems | 1
  Tumor Assessment Week 165: Moderate Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Moderate Problems | 1
  Tumor Assessment Week 165: Invalid Response: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Invalid Response | 1
  Tumor Assessment Week 174: No Problem: number analyzed (Participants) | 10
  Tumor Assessment Week 174: No Problem | 9
  Tumor Assessment Week 174: Slight Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 174: Slight Problems | 1
  Tumor Assessment Week 183: No Problem: number analyzed (Participants) | 3
  Tumor Assessment Week 183: No Problem | 1
  Tumor Assessment Week 183: Slight Problems: number analyzed (Participants) | 3
  Tumor Assessment Week 183: Slight Problems | 2

7. Secondary Outcome: EQ-5D-5L Questionnaire - Usual Activities Item
Description: The EQ-5D-5L was a self-reported health status questionnaire that consisted of six questions used to calculate a health utility score for use in health economic analysis. The EQ-5D-5L has two components: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, as well as a VAS that measures health state. Each item was rated from 1 (no problems) to 5 (extreme problems). Categories with non-zero values are reported here. Number of participants who rated the usual activities item ranging from 1-5 are reported. Participants who had a invalid response were presented under the category 'Invalid Response'.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Participants
  Baseline: No Problem: number analyzed (Participants) | 597
  Baseline: No Problem | 297
  Baseline: Slight Problem: number analyzed (Participants) | 597
  Baseline: Slight Problem | 164
  Baseline: Moderate Problems: number analyzed (Participants) | 597
  Baseline: Moderate Problems | 99
  Baseline: Severe Problems: number analyzed (Participants) | 597
  Baseline: Severe Problems | 16
  Baseline: Extreme Problems: number analyzed (Participants) | 597
  Baseline: Extreme Problems | 21
  Cycle 2 Day 1: No Problem: number analyzed (Participants) | 534
  Cycle 2 Day 1: No Problem | 257
  Cycle 2 Day 1: Slight Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Slight Problems | 152
  Cycle 2 Day 1: Moderate Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Moderate Problems | 85
  Cycle 2 Day 1: Severe Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Severe Problems | 24
  Cycle 2 Day 1: Extreme Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Extreme Problems | 16
  Tumor Assessment Week 006: No Problem: number analyzed (Participants) | 438
  Tumor Assessment Week 006: No Problem | 221
  Tumor Assessment Week 006: Slight Problems: number analyzed (Participants) | 438
  Tumor Assessment Week 006: Slight Problems | 121
  Tumor Assessment Week 006: Moderate Problems: number analyzed (Participants) | 438
  Tumor Assessment Week 006: Moderate Problems | 69
  Tumor Assessment Week 006: Severe Problems: number analyzed (Participants) | 438
  Tumor Assessment Week 006: Severe Problems | 14
  Tumor Assessment Week 006: Extreme Problems: number analyzed (Participants) | 438
  Tumor Assessment Week 006: Extreme Problems | 13
  Tumor Assessment Week 012: No Problem: number analyzed (Participants) | 323
  Tumor Assessment Week 012: No Problem | 175
  Tumor Assessment Week 012: Slight Problems: number analyzed (Participants) | 323
  Tumor Assessment Week 012: Slight Problems | 83
  Tumor Assessment Week 012: Moderate Problems: number analyzed (Participants) | 323
  Tumor Assessment Week 012: Moderate Problems | 47
  Tumor Assessment Week 012: Severe Problems: number analyzed (Participants) | 323
  Tumor Assessment Week 012: Severe Problems | 10
  Tumor Assessment Week 012: Extreme Problems: number analyzed (Participants) | 323
  Tumor Assessment Week 012: Extreme Problems | 8
  Tumor Assessment Week 018: No Problem: number analyzed (Participants) | 260
  Tumor Assessment Week 018: No Problem | 143
  Tumor Assessment Week 018: Slight Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Slight Problems | 80
  Tumor Assessment Week 018: Moderate Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Moderate Problems | 29
  Tumor Assessment Week 018: Severe Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Severe Problems | 3
  Tumor Assessment Week 018: Extreme Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Extreme Problems | 5
  Tumor Assessment Week 024: No Problem: number analyzed (Participants) | 220
  Tumor Assessment Week 024: No Problem | 134
  Tumor Assessment Week 024: Slight Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Slight Problems | 56
  Tumor Assessment Week 024: Moderate Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Moderate Problems | 22
  Tumor Assessment Week 024: Severe Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Severe Problems | 1
  Tumor Assessment Week 024: Extreme Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Extreme Problems | 6
  Tumor Assessment Week 024: Invalid Response: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Invalid Response | 1
  Tumor Assessment Week 030: No Problem: number analyzed (Participants) | 184
  Tumor Assessment Week 030: No Problem | 124
  Tumor Assessment Week 030: Slight Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Slight Problems | 43
  Tumor Assessment Week 030: Moderate Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Moderate Problems | 9
  Tumor Assessment Week 030: Severe Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Severe Problems | 5
  Tumor Assessment Week 030: Extreme Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Extreme Problems | 3
  Tumor Assessment Week 036: No Problem: number analyzed (Participants) | 162
  Tumor Assessment Week 036: No Problem | 107
  Tumor Assessment Week 036: Slight Problems: number analyzed (Participants) | 162
  Tumor Assessment Week 036: Slight Problems | 38
  Tumor Assessment Week 036: Moderate Problems: number analyzed (Participants) | 162
  Tumor Assessment Week 036: Moderate Problems | 13
  Tumor Assessment Week 036: Severe Problems: number analyzed (Participants) | 162
  Tumor Assessment Week 036: Severe Problems | 3
  Tumor Assessment Week 036: Extreme Problems: number analyzed (Participants) | 162
  Tumor Assessment Week 036: Extreme Problems | 1
  Tumor Assessment Week 042: No Problem: number analyzed (Participants) | 145
  Tumor Assessment Week 042: No Problem | 97
  Tumor Assessment Week 042: Slight Problems: number analyzed (Participants) | 145
  Tumor Assessment Week 042: Slight Problems | 32
  Tumor Assessment Week 042: Moderate Problems: number analyzed (Participants) | 145
  Tumor Assessment Week 042: Moderate Problems | 11
  Tumor Assessment Week 042: Severe Problems: number analyzed (Participants) | 145
  Tumor Assessment Week 042: Severe Problems | 3
  Tumor Assessment Week 042: Extreme Problems: number analyzed (Participants) | 145
  Tumor Assessment Week 042: Extreme Problems | 2
  Tumor Assessment Week 048: No Problem: number analyzed (Participants) | 127
  Tumor Assessment Week 048: No Problem | 81
  Tumor Assessment Week 048: Slight Problems: number analyzed (Participants) | 127
  Tumor Assessment Week 048: Slight Problems | 31
  Tumor Assessment Week 048: Moderate Problems: number analyzed (Participants) | 127
  Tumor Assessment Week 048: Moderate Problems | 8
  Tumor Assessment Week 048: Severe Problems: number analyzed (Participants) | 127
  Tumor Assessment Week 048: Severe Problems | 5
  Tumor Assessment Week 048: Extreme Problems: number analyzed (Participants) | 127
  Tumor Assessment Week 048: Extreme Problems | 1
  Tumor Assessment Week 048: Invalid Response: number analyzed (Participants) | 127
  Tumor Assessment Week 048: Invalid Response | 1
  Tumor Assessment Week 054: No Problem: number analyzed (Participants) | 23
  Tumor Assessment Week 054: No Problem | 10
  Tumor Assessment Week 054: Slight Problems: number analyzed (Participants) | 23
  Tumor Assessment Week 054: Slight Problems | 8
  Tumor Assessment Week 054: Moderate Problems: number analyzed (Participants) | 23
  Tumor Assessment Week 054: Moderate Problems | 3
  Tumor Assessment Week 054: Severe Problems: number analyzed (Participants) | 23
  Tumor Assessment Week 054: Severe Problems | 1
  Tumor Assessment Week 054: Extreme Problems: number analyzed (Participants) | 23
  Tumor Assessment Week 054: Extreme Problems | 1
  Tumor Assessment Week 057: No Problem: number analyzed (Participants) | 97
  Tumor Assessment Week 057: No Problem | 61
  Tumor Assessment Week 057: Slight Problems: number analyzed (Participants) | 97
  Tumor Assessment Week 057: Slight Problems | 23
  Tumor Assessment Week 057: Moderate Problems: number analyzed (Participants) | 97
  Tumor Assessment Week 057: Moderate Problems | 7
  Tumor Assessment Week 057: Severe Problems: number analyzed (Participants) | 97
  Tumor Assessment Week 057: Severe Problems | 1
  Tumor Assessment Week 057: Extreme Problems: number analyzed (Participants) | 97
  Tumor Assessment Week 057: Extreme Problems | 4
  Tumor Assessment Week 057: Invalid Response: number analyzed (Participants) | 97
  Tumor Assessment Week 057: Invalid Response | 1
  Tumor Assessment Week 060: No Problem: number analyzed (Participants) | 17
  Tumor Assessment Week 060: No Problem | 12
  Tumor Assessment Week 060: Slight Problems: number analyzed (Participants) | 17
  Tumor Assessment Week 060: Slight Problems | 3
  Tumor Assessment Week 060: Moderate Problems: number analyzed (Participants) | 17
  Tumor Assessment Week 060: Moderate Problems | 1
  Tumor Assessment Week 060: Extreme Problems: number analyzed (Participants) | 17
  Tumor Assessment Week 060: Extreme Problems | 1
  Tumor Assessment Week 066: No Problem: number analyzed (Participants) | 88
  Tumor Assessment Week 066: No Problem | 58
  Tumor Assessment Week 066: Slight Problems: number analyzed (Participants) | 88
  Tumor Assessment Week 066: Slight Problems | 19
  Tumor Assessment Week 066: Moderate Problems: number analyzed (Participants) | 88
  Tumor Assessment Week 066: Moderate Problems | 7
  Tumor Assessment Week 066: Severe Problems: number analyzed (Participants) | 88
  Tumor Assessment Week 066: Severe Problems | 4
  Tumor Assessment Week 072: No Problem: number analyzed (Participants) | 13
  Tumor Assessment Week 072: No Problem | 7
  Tumor Assessment Week 072: Slight Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 072: Slight Problems | 4
  Tumor Assessment Week 072: Moderate Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 072: Moderate Problems | 1
  Tumor Assessment Week 072: Severe Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 072: Severe Problems | 1
  Tumor Assessment Week 075: No Problem: number analyzed (Participants) | 73
  Tumor Assessment Week 075: No Problem | 47
  Tumor Assessment Week 075: Slight Problems: number analyzed (Participants) | 73
  Tumor Assessment Week 075: Slight Problems | 21
  Tumor Assessment Week 075: Moderate Problems: number analyzed (Participants) | 73
  Tumor Assessment Week 075: Moderate Problems | 5
  Tumor Assessment Week 078: No Problem: number analyzed (Participants) | 10
  Tumor Assessment Week 078: No Problem | 6
  Tumor Assessment Week 078: Slight Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 078: Slight Problems | 2
  Tumor Assessment Week 078: Moderate Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 078: Moderate Problems | 1
  Tumor Assessment Week 078: Severe Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 078: Severe Problems | 1
  Tumor Assessment Week 084: No Problem: number analyzed (Participants) | 67
  Tumor Assessment Week 084: No Problem | 46
  Tumor Assessment Week 084: Slight Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Slight Problems | 12
  Tumor Assessment Week 084: Moderate Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Moderate Problems | 6
  Tumor Assessment Week 084: Severe Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Severe Problems | 1
  Tumor Assessment Week 084: Extreme Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Extreme Problems | 2
  Tumor Assessment Week 090: No Problem: number analyzed (Participants) | 10
  Tumor Assessment Week 090: No Problem | 6
  Tumor Assessment Week 090: Slight Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 090: Slight Problems | 3
  Tumor Assessment Week 090: Severe Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 090: Severe Problems | 1
  Tumor Assessment Week 093: No Problem: number analyzed (Participants) | 53
  Tumor Assessment Week 093: No Problem | 36
  Tumor Assessment Week 093: Slight Problems: number analyzed (Participants) | 53
  Tumor Assessment Week 093: Slight Problems | 12
  Tumor Assessment Week 093: Moderate Problems: number analyzed (Participants) | 53
  Tumor Assessment Week 093: Moderate Problems | 4
  Tumor Assessment Week 093: Extreme Problems: number analyzed (Participants) | 53
  Tumor Assessment Week 093: Extreme Problems | 1
  Tumor Assessment Week 096: No Problem: number analyzed (Participants) | 7
  Tumor Assessment Week 096: No Problem | 5
  Tumor Assessment Week 096: Slight Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 096: Slight Problems | 1
  Tumor Assessment Week 096: Severe Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 096: Severe Problems | 1
  Tumor Assessment Week 102: No Problem: number analyzed (Participants) | 55
  Tumor Assessment Week 102: No Problem | 36
  Tumor Assessment Week 102: Slight Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Slight Problems | 13
  Tumor Assessment Week 102: Moderate Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Moderate Problems | 3
  Tumor Assessment Week 102: Severe Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Severe Problems | 2
  Tumor Assessment Week 102: Extreme Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Extreme Problems | 1
  Tumor Assessment Week 108: No Problem: number analyzed (Participants) | 7
  Tumor Assessment Week 108: No Problem | 3
  Tumor Assessment Week 108: Slight Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 108: Slight Problems | 4
  Tumor Assessment Week 111: No Problem: number analyzed (Participants) | 41
  Tumor Assessment Week 111: No Problem | 25
  Tumor Assessment Week 111: Slight Problems: number analyzed (Participants) | 41
  Tumor Assessment Week 111: Slight Problems | 12
  Tumor Assessment Week 111: Moderate Problems: number analyzed (Participants) | 41
  Tumor Assessment Week 111: Moderate Problems | 3
  Tumor Assessment Week 111: Extreme Problems: number analyzed (Participants) | 41
  Tumor Assessment Week 111: Extreme Problems | 1
  Tumor Assessment Week 114: Slight Problems: number analyzed (Participants) | 2
  Tumor Assessment Week 114: Slight Problems | 1
  Tumor Assessment Week 114: Moderate Problems: number analyzed (Participants) | 2
  Tumor Assessment Week 114: Moderate Problems | 1
  Tumor Assessment Week 120: No Problem: number analyzed (Participants) | 38
  Tumor Assessment Week 120: No Problem | 27
  Tumor Assessment Week 120: Slight Problems: number analyzed (Participants) | 38
  Tumor Assessment Week 120: Slight Problems | 10
  Tumor Assessment Week 120: Extreme Problems: number analyzed (Participants) | 38
  Tumor Assessment Week 120: Extreme Problems | 1
  Tumor Assessment Week 126: No Problem: number analyzed (Participants) | 4
  Tumor Assessment Week 126: No Problem | 1
  Tumor Assessment Week 126: Slight Problems: number analyzed (Participants) | 4
  Tumor Assessment Week 126: Slight Problems | 3
  Tumor Assessment Week 129: No Problem: number analyzed (Participants) | 32
  Tumor Assessment Week 129: No Problem | 22
  Tumor Assessment Week 129: Slight Problems: number analyzed (Participants) | 32
  Tumor Assessment Week 129: Slight Problems | 9
  Tumor Assessment Week 129: Extreme Problems: number analyzed (Participants) | 32
  Tumor Assessment Week 129: Extreme Problems | 1
  Tumor Assessment Week 132: No Problem: number analyzed (Participants) | 2
  Tumor Assessment Week 132: No Problem | 1
  Tumor Assessment Week 132: Moderate Problems: number analyzed (Participants) | 2
  Tumor Assessment Week 132: Moderate Problems | 1
  Tumor Assessment Week 138: No Problem: number analyzed (Participants) | 28
  Tumor Assessment Week 138: No Problem | 16
  Tumor Assessment Week 138: Slight Problems: number analyzed (Participants) | 28
  Tumor Assessment Week 138: Slight Problems | 10
  Tumor Assessment Week 138: Moderate Problems: number analyzed (Participants) | 28
  Tumor Assessment Week 138: Moderate Problems | 2
  Tumor Assessment Week 144: No Problem: number analyzed (Participants) | 1
  Tumor Assessment Week 144: No Problem | 1
  Tumor Assessment Week 147: No Problem: number analyzed (Participants) | 21
  Tumor Assessment Week 147: No Problem | 12
  Tumor Assessment Week 147: Slight Problems: number analyzed (Participants) | 21
  Tumor Assessment Week 147: Slight Problems | 7
  Tumor Assessment Week 147: Moderate Problems: number analyzed (Participants) | 21
  Tumor Assessment Week 147: Moderate Problems | 2
  Tumor Assessment Week 156: No Problem: number analyzed (Participants) | 15
  Tumor Assessment Week 156: No Problem | 9
  Tumor Assessment Week 156: Slight Problems: number analyzed (Participants) | 15
  Tumor Assessment Week 156: Slight Problems | 5
  Tumor Assessment Week 156: Extreme Problems: number analyzed (Participants) | 15
  Tumor Assessment Week 156: Extreme Problems | 1
  Tumor Assessment Week 165: No Problem: number analyzed (Participants) | 13
  Tumor Assessment Week 165: No Problem | 6
  Tumor Assessment Week 165: Slight Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Slight Problems | 4
  Tumor Assessment Week 165: Moderate Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Moderate Problems | 1
  Tumor Assessment Week 165: Extreme Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Extreme Problems | 1
  Tumor Assessment Week 165: Invalid Response: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Invalid Response | 1
  Tumor Assessment Week 174: No Problem: number analyzed (Participants) | 10
  Tumor Assessment Week 174: No Problem | 8
  Tumor Assessment Week 174: Slight Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 174: Slight Problems | 2
  Tumor Assessment Week 183: Slight Problems: number analyzed (Participants) | 3
  Tumor Assessment Week 183: Slight Problems | 3

8. Secondary Outcome: EQ-5D-5L Questionnaire - Pain/Discomfort Item
Description: The EQ-5D-5L was a self-reported health status questionnaire that consisted of six questions used to calculate a health utility score for use in health economic analysis. The EQ-5D-5L has two components: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, as well as a VAS that measures health state. Each item was rated from 1 (no problems) to 5 (extreme problems). Categories with non-zero values are reported here. Number of participants who rated the pain/discomfort item ranging from 1-5 are reported. Participants who had a invalid response were presented under the category 'Invalid Response'.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Participants
  Baseline: No Problem: number analyzed (Participants) | 597
  Baseline: No Problem | 206
  Baseline: Slight Problem: number analyzed (Participants) | 597
  Baseline: Slight Problem | 216
  Baseline: Moderate Problems: number analyzed (Participants) | 597
  Baseline: Moderate Problems | 129
  Baseline: Severe Problems: number analyzed (Participants) | 597
  Baseline: Severe Problems | 38
  Baseline: Extreme Problems: number analyzed (Participants) | 597
  Baseline: Extreme Problems | 7
  Baseline: Invalid Response: number analyzed (Participants) | 597
  Baseline: Invalid Response | 1
  Cycle 2 Day 1: No Problem: number analyzed (Participants) | 534
  Cycle 2 Day 1: No Problem | 212
  Cycle 2 Day 1: Slight Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Slight Problems | 165
  Cycle 2 Day 1: Moderate Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Moderate Problems | 117
  Cycle 2 Day 1: Severe Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Severe Problems | 34
  Cycle 2 Day 1: Extreme Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Extreme Problems | 6
  Tumor Assessment Week 006: No Problem: number analyzed (Participants) | 437
  Tumor Assessment Week 006: No Problem | 165
  Tumor Assessment Week 006: Slight Problems: number analyzed (Participants) | 437
  Tumor Assessment Week 006: Slight Problems | 143
  Tumor Assessment Week 006: Moderate Problems: number analyzed (Participants) | 437
  Tumor Assessment Week 006: Moderate Problems | 93
  Tumor Assessment Week 006: Severe Problems: number analyzed (Participants) | 437
  Tumor Assessment Week 006: Severe Problems | 31
  Tumor Assessment Week 006: Extreme Problems: number analyzed (Participants) | 437
  Tumor Assessment Week 006: Extreme Problems | 5
  Tumor Assessment Week 012: No Problem: number analyzed (Participants) | 322
  Tumor Assessment Week 012: No Problem | 125
  Tumor Assessment Week 012: Slight Problems: number analyzed (Participants) | 322
  Tumor Assessment Week 012: Slight Problems | 116
  Tumor Assessment Week 012: Moderate Problems: number analyzed (Participants) | 322
  Tumor Assessment Week 012: Moderate Problems | 61
  Tumor Assessment Week 012: Severe Problems: number analyzed (Participants) | 322
  Tumor Assessment Week 012: Severe Problems | 16
  Tumor Assessment Week 012: Extreme Problems: number analyzed (Participants) | 322
  Tumor Assessment Week 012: Extreme Problems | 4
  Tumor Assessment Week 018: No Problem: number analyzed (Participants) | 260
  Tumor Assessment Week 018: No Problem | 123
  Tumor Assessment Week 018: Slight Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Slight Problems | 88
  Tumor Assessment Week 018: Moderate Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Moderate Problems | 32
  Tumor Assessment Week 018: Severe Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Severe Problems | 15
  Tumor Assessment Week 018: Extreme Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Extreme Problems | 1
  Tumor Assessment Week 018: Invalid Response: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Invalid Response | 1
  Tumor Assessment Week 024: No Problem: number analyzed (Participants) | 220
  Tumor Assessment Week 024: No Problem | 101
  Tumor Assessment Week 024: Slight Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Slight Problems | 74
  Tumor Assessment Week 024: Moderate Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Moderate Problems | 33
  Tumor Assessment Week 024: Severe Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Severe Problems | 10
  Tumor Assessment Week 024: Extreme Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Extreme Problems | 1
  Tumor Assessment Week 024: Invalid Response: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Invalid Response | 1
  Tumor Assessment Week 030: No Problem: number analyzed (Participants) | 184
  Tumor Assessment Week 030: No Problem | 89
  Tumor Assessment Week 030: Slight Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Slight Problems | 64
  Tumor Assessment Week 030: Moderate Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Moderate Problems | 25
  Tumor Assessment Week 030: Severe Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Severe Problems | 6
  Tumor Assessment Week 036: No Problem: number analyzed (Participants) | 162
  Tumor Assessment Week 036: No Problem | 85
  Tumor Assessment Week 036: Slight Problems: number analyzed (Participants) | 162
  Tumor Assessment Week 036: Slight Problems | 51
  Tumor Assessment Week 036: Moderate Problems: number analyzed (Participants) | 162
  Tumor Assessment Week 036: Moderate Problems | 19
  Tumor Assessment Week 036: Severe Problems: number analyzed (Participants) | 162
  Tumor Assessment Week 036: Severe Problems | 6
  Tumor Assessment Week 036: Extreme Problems: number analyzed (Participants) | 162
  Tumor Assessment Week 036: Extreme Problems | 1
  Tumor Assessment Week 042: No Problem: number analyzed (Participants) | 145
  Tumor Assessment Week 042: No Problem | 68
  Tumor Assessment Week 042: Slight Problems: number analyzed (Participants) | 145
  Tumor Assessment Week 042: Slight Problems | 51
  Tumor Assessment Week 042: Moderate Problems: number analyzed (Participants) | 145
  Tumor Assessment Week 042: Moderate Problems | 19
  Tumor Assessment Week 042: Severe Problems: number analyzed (Participants) | 145
  Tumor Assessment Week 042: Severe Problems | 6
  Tumor Assessment Week 042: Extreme Problems: number analyzed (Participants) | 145
  Tumor Assessment Week 042: Extreme Problems | 1
  Tumor Assessment Week 048: No Problem: number analyzed (Participants) | 127
  Tumor Assessment Week 048: No Problem | 64
  Tumor Assessment Week 048: Slight Problems: number analyzed (Participants) | 127
  Tumor Assessment Week 048: Slight Problems | 41
  Tumor Assessment Week 048: Moderate Problems: number analyzed (Participants) | 127
  Tumor Assessment Week 048: Moderate Problems | 15
  Tumor Assessment Week 048: Severe Problems: number analyzed (Participants) | 127
  Tumor Assessment Week 048: Severe Problems | 5
  Tumor Assessment Week 048: Extreme Problems: number analyzed (Participants) | 127
  Tumor Assessment Week 048: Extreme Problems | 2
  Tumor Assessment Week 054: No Problem: number analyzed (Participants) | 23
  Tumor Assessment Week 054: No Problem | 9
  Tumor Assessment Week 054: Slight Problems: number analyzed (Participants) | 23
  Tumor Assessment Week 054: Slight Problems | 10
  Tumor Assessment Week 054: Moderate Problems: number analyzed (Participants) | 23
  Tumor Assessment Week 054: Moderate Problems | 4
  Tumor Assessment Week 057: No Problem: number analyzed (Participants) | 97
  Tumor Assessment Week 057: No Problem | 53
  Tumor Assessment Week 057: Slight Problems: number analyzed (Participants) | 97
  Tumor Assessment Week 057: Slight Problems | 27
  Tumor Assessment Week 057: Moderate Problems: number analyzed (Participants) | 97
  Tumor Assessment Week 057: Moderate Problems | 12
  Tumor Assessment Week 057: Severe Problems: number analyzed (Participants) | 97
  Tumor Assessment Week 057: Severe Problems | 5
  Tumor Assessment Week 060: No Problem: number analyzed (Participants) | 17
  Tumor Assessment Week 060: No Problem | 12
  Tumor Assessment Week 060: Slight Problems: number analyzed (Participants) | 17
  Tumor Assessment Week 060: Slight Problems | 3
  Tumor Assessment Week 060: Moderate Problems: number analyzed (Participants) | 17
  Tumor Assessment Week 060: Moderate Problems | 2
  Tumor Assessment Week 066: No Problem: number analyzed (Participants) | 88
  Tumor Assessment Week 066: No Problem | 48
  Tumor Assessment Week 066: Slight Problems: number analyzed (Participants) | 88
  Tumor Assessment Week 066: Slight Problems | 27
  Tumor Assessment Week 066: Moderate Problems: number analyzed (Participants) | 88
  Tumor Assessment Week 066: Moderate Problems | 8
  Tumor Assessment Week 066: Severe Problems: number analyzed (Participants) | 88
  Tumor Assessment Week 066: Severe Problems | 5
  Tumor Assessment Week 072: No Problem: number analyzed (Participants) | 13
  Tumor Assessment Week 072: No Problem | 7
  Tumor Assessment Week 072: Slight Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 072: Slight Problems | 5
  Tumor Assessment Week 072: Moderate Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 072: Moderate Problems | 1
  Tumor Assessment Week 075: No Problem: number analyzed (Participants) | 73
  Tumor Assessment Week 075: No Problem | 45
  Tumor Assessment Week 075: Slight Problems: number analyzed (Participants) | 73
  Tumor Assessment Week 075: Slight Problems | 19
  Tumor Assessment Week 075: Moderate Problems: number analyzed (Participants) | 73
  Tumor Assessment Week 075: Moderate Problems | 8
  Tumor Assessment Week 075: Extreme Problems: number analyzed (Participants) | 73
  Tumor Assessment Week 075: Extreme Problems | 1
  Tumor Assessment Week 078: No Problem: number analyzed (Participants) | 10
  Tumor Assessment Week 078: No Problem | 6
  Tumor Assessment Week 078: Slight Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 078: Slight Problems | 3
  Tumor Assessment Week 078: Severe Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 078: Severe Problems | 1
  Tumor Assessment Week 084: No Problem: number analyzed (Participants) | 67
  Tumor Assessment Week 084: No Problem | 41
  Tumor Assessment Week 084: Slight Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Slight Problems | 18
  Tumor Assessment Week 084: Moderate Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Moderate Problems | 5
  Tumor Assessment Week 084: Severe Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Severe Problems | 3
  Tumor Assessment Week 090: No Problem: number analyzed (Participants) | 10
  Tumor Assessment Week 090: No Problem | 8
  Tumor Assessment Week 090: Slight Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 090: Slight Problems | 1
  Tumor Assessment Week 090: Severe Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 090: Severe Problems | 1
  Tumor Assessment Week 093: No Problem: number analyzed (Participants) | 53
  Tumor Assessment Week 093: No Problem | 34
  Tumor Assessment Week 093: Slight Problems: number analyzed (Participants) | 53
  Tumor Assessment Week 093: Slight Problems | 14
  Tumor Assessment Week 093: Moderate Problems: number analyzed (Participants) | 53
  Tumor Assessment Week 093: Moderate Problems | 2
  Tumor Assessment Week 093: Severe Problems: number analyzed (Participants) | 53
  Tumor Assessment Week 093: Severe Problems | 3
  Tumor Assessment Week 096: No Problem: number analyzed (Participants) | 7
  Tumor Assessment Week 096: No Problem | 4
  Tumor Assessment Week 096: Slight Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 096: Slight Problems | 2
  Tumor Assessment Week 096: Severe Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 096: Severe Problems | 1
  Tumor Assessment Week 102: No Problem: number analyzed (Participants) | 55
  Tumor Assessment Week 102: No Problem | 33
  Tumor Assessment Week 102: Slight Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Slight Problems | 16
  Tumor Assessment Week 102: Moderate Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Moderate Problems | 4
  Tumor Assessment Week 102: Severe Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Severe Problems | 2
  Tumor Assessment Week 108: No Problem: number analyzed (Participants) | 7
  Tumor Assessment Week 108: No Problem | 4
  Tumor Assessment Week 108: Slight Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 108: Slight Problems | 3
  Tumor Assessment Week 111: No Problem: number analyzed (Participants) | 41
  Tumor Assessment Week 111: No Problem | 21
  Tumor Assessment Week 111: Slight Problems: number analyzed (Participants) | 41
  Tumor Assessment Week 111: Slight Problems | 17
  Tumor Assessment Week 111: Moderate Problems: number analyzed (Participants) | 41
  Tumor Assessment Week 111: Moderate Problems | 2
  Tumor Assessment Week 111: Extreme Problems: number analyzed (Participants) | 41
  Tumor Assessment Week 111: Extreme Problems | 1
  Tumor Assessment Week 114: Slight Problems: number analyzed (Participants) | 2
  Tumor Assessment Week 114: Slight Problems | 1
  Tumor Assessment Week 114: Moderate Problems: number analyzed (Participants) | 2
  Tumor Assessment Week 114: Moderate Problems | 1
  Tumor Assessment Week 120: No Problem: number analyzed (Participants) | 38
  Tumor Assessment Week 120: No Problem | 20
  Tumor Assessment Week 120: Slight Problems: number analyzed (Participants) | 38
  Tumor Assessment Week 120: Slight Problems | 14
  Tumor Assessment Week 120: Moderate Problems: number analyzed (Participants) | 38
  Tumor Assessment Week 120: Moderate Problems | 4
  Tumor Assessment Week 126: No Problem: number analyzed (Participants) | 4
  Tumor Assessment Week 126: No Problem | 1
  Tumor Assessment Week 126: Slight Problems: number analyzed (Participants) | 4
  Tumor Assessment Week 126: Slight Problems | 3
  Tumor Assessment Week 129: No Problem: number analyzed (Participants) | 32
  Tumor Assessment Week 129: No Problem | 17
  Tumor Assessment Week 129: Slight Problems: number analyzed (Participants) | 32
  Tumor Assessment Week 129: Slight Problems | 13
  Tumor Assessment Week 129: Moderate Problems: number analyzed (Participants) | 32
  Tumor Assessment Week 129: Moderate Problems | 1
  Tumor Assessment Week 129: Severe Problems: number analyzed (Participants) | 32
  Tumor Assessment Week 129: Severe Problems | 1
  Tumor Assessment Week 132: No Problem: number analyzed (Participants) | 2
  Tumor Assessment Week 132: No Problem | 1
  Tumor Assessment Week 132: Slight Problems: number analyzed (Participants) | 2
  Tumor Assessment Week 132: Slight Problems | 1
  Tumor Assessment Week 138: No Problem: number analyzed (Participants) | 28
  Tumor Assessment Week 138: No Problem | 15
  Tumor Assessment Week 138: Slight Problems: number analyzed (Participants) | 28
  Tumor Assessment Week 138: Slight Problems | 10
  Tumor Assessment Week 138: Moderate Problems: number analyzed (Participants) | 28
  Tumor Assessment Week 138: Moderate Problems | 2
  Tumor Assessment Week 138: Severe Problems: number analyzed (Participants) | 28
  Tumor Assessment Week 138: Severe Problems | 1
  Tumor Assessment Week 144: No Problem: number analyzed (Participants) | 1
  Tumor Assessment Week 144: No Problem | 1
  Tumor Assessment Week 147: No Problem: number analyzed (Participants) | 21
  Tumor Assessment Week 147: No Problem | 11
  Tumor Assessment Week 147: Slight Problems: number analyzed (Participants) | 21
  Tumor Assessment Week 147: Slight Problems | 8
  Tumor Assessment Week 147: Moderate Problems: number analyzed (Participants) | 21
  Tumor Assessment Week 147: Moderate Problems | 2
  Tumor Assessment Week 156: No Problem: number analyzed (Participants) | 15
  Tumor Assessment Week 156: No Problem | 8
  Tumor Assessment Week 156: Slight Problems: number analyzed (Participants) | 15
  Tumor Assessment Week 156: Slight Problems | 4
  Tumor Assessment Week 156: Moderate Problems: number analyzed (Participants) | 15
  Tumor Assessment Week 156: Moderate Problems | 3
  Tumor Assessment Week 165: No Problem: number analyzed (Participants) | 13
  Tumor Assessment Week 165: No Problem | 4
  Tumor Assessment Week 165: Slight Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Slight Problems | 5
  Tumor Assessment Week 165: Moderate Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Moderate Problems | 2
  Tumor Assessment Week 165: Severe Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Severe Problems | 1
  Tumor Assessment Week 165: Invalid Response: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Invalid Response | 1
  Tumor Assessment Week 174: No Problem: number analyzed (Participants) | 10
  Tumor Assessment Week 174: No Problem | 5
  Tumor Assessment Week 174: Slight Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 174: Slight Problems | 3
  Tumor Assessment Week 174: Moderate Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 174: Moderate Problems | 2
  Tumor Assessment Week 183: Slight Problems: number analyzed (Participants) | 3
  Tumor Assessment Week 183: Slight Problems | 2
  Tumor Assessment Week 183: Moderate Problems: number analyzed (Participants) | 3
  Tumor Assessment Week 183: Moderate Problems | 1

9. Secondary Outcome: EQ-5D-5L Questionnaire - Anxiety/Depression Item
Description: The EQ-5D-5L was a self-reported health status questionnaire that consisted of six questions used to calculate a health utility score for use in health economic analysis. The EQ-5D-5L has two components: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, as well as a VAS that measures health state. Each item was rated from 1 (no problems) to 5 (extreme problems). Categories with non-zero values are reported here. Number of participants who rated the anxiety/depression item ranging from 1-5 are reported. Participants who had a invalid response were presented under the category 'Invalid Response'.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Participants
  Baseline: No Problem: number analyzed (Participants) | 597
  Baseline: No Problem | 334
  Baseline: Slight Problem: number analyzed (Participants) | 597
  Baseline: Slight Problem | 163
  Baseline: Moderate Problems: number analyzed (Participants) | 597
  Baseline: Moderate Problems | 83
  Baseline: Severe Problems: number analyzed (Participants) | 597
  Baseline: Severe Problems | 13
  Baseline: Extreme Problems: number analyzed (Participants) | 597
  Baseline: Extreme Problems | 3
  Baseline: Invalid Response: number analyzed (Participants) | 597
  Baseline: Invalid Response | 1
  Cycle 2 Day 1: No Problem: number analyzed (Participants) | 534
  Cycle 2 Day 1: No Problem | 296
  Cycle 2 Day 1: Slight Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Slight Problems | 157
  Cycle 2 Day 1: Moderate Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Moderate Problems | 66
  Cycle 2 Day 1: Severe Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Severe Problems | 9
  Cycle 2 Day 1: Extreme Problems: number analyzed (Participants) | 534
  Cycle 2 Day 1: Extreme Problems | 4
  Cycle 2 Day 1: Invalid Response: number analyzed (Participants) | 534
  Cycle 2 Day 1: Invalid Response | 2
  Tumor Assessment Week 006: No Problem: number analyzed (Participants) | 437
  Tumor Assessment Week 006: No Problem | 267
  Tumor Assessment Week 006: Slight Problems: number analyzed (Participants) | 437
  Tumor Assessment Week 006: Slight Problems | 109
  Tumor Assessment Week 006: Moderate Problems: number analyzed (Participants) | 437
  Tumor Assessment Week 006: Moderate Problems | 49
  Tumor Assessment Week 006: Severe Problems: number analyzed (Participants) | 437
  Tumor Assessment Week 006: Severe Problems | 10
  Tumor Assessment Week 006: Extreme Problems: number analyzed (Participants) | 437
  Tumor Assessment Week 006: Extreme Problems | 2
  Tumor Assessment Week 012: No Problem: number analyzed (Participants) | 322
  Tumor Assessment Week 012: No Problem | 190
  Tumor Assessment Week 012: Slight Problems: number analyzed (Participants) | 322
  Tumor Assessment Week 012: Slight Problems | 102
  Tumor Assessment Week 012: Moderate Problems: number analyzed (Participants) | 322
  Tumor Assessment Week 012: Moderate Problems | 20
  Tumor Assessment Week 012: Severe Problems: number analyzed (Participants) | 322
  Tumor Assessment Week 012: Severe Problems | 8
  Tumor Assessment Week 012: Extreme Problems: number analyzed (Participants) | 322
  Tumor Assessment Week 012: Extreme Problems | 2
  Tumor Assessment Week 018: No Problem: number analyzed (Participants) | 260
  Tumor Assessment Week 018: No Problem | 167
  Tumor Assessment Week 018: Slight Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Slight Problems | 66
  Tumor Assessment Week 018: Moderate Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Moderate Problems | 22
  Tumor Assessment Week 018: Severe Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Severe Problems | 4
  Tumor Assessment Week 018: Invalid Response: number analyzed (Participants) | 260
  Tumor Assessment Week 018: Invalid Response | 1
  Tumor Assessment Week 024: No Problem: number analyzed (Participants) | 220
  Tumor Assessment Week 024: No Problem | 140
  Tumor Assessment Week 024: Slight Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Slight Problems | 62
  Tumor Assessment Week 024: Moderate Problems: number analyzed (Participants) | 220
  Tumor Assessment Week 024: Moderate Problems | 13
  Tumor Assessment Week 024: Severe Problems: number analyzed (Participants) | 260
  Tumor Assessment Week 024: Severe Problems | 5
  Tumor Assessment Week 030: No Problem: number analyzed (Participants) | 184
  Tumor Assessment Week 030: No Problem | 116
  Tumor Assessment Week 030: Slight Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Slight Problems | 56
  Tumor Assessment Week 030: Moderate Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Moderate Problems | 11
  Tumor Assessment Week 030: Severe Problems: number analyzed (Participants) | 184
  Tumor Assessment Week 030: Severe Problems | 1
  Tumor Assessment Week 036: No Problem: number analyzed (Participants) | 162
  Tumor Assessment Week 036: No Problem | 105
  Tumor Assessment Week 036: Slight Problems: number analyzed (Participants) | 162
  Tumor Assessment Week 036: Slight Problems | 46
  Tumor Assessment Week 036: Moderate Problems: number analyzed (Participants) | 162
  Tumor Assessment Week 036: Moderate Problems | 9
  Tumor Assessment Week 036: Severe Problems: number analyzed (Participants) | 162
  Tumor Assessment Week 036: Severe Problems | 2
  Tumor Assessment Week 042: No Problem: number analyzed (Participants) | 145
  Tumor Assessment Week 042: No Problem | 90
  Tumor Assessment Week 042: Slight Problems: number analyzed (Participants) | 145
  Tumor Assessment Week 042: Slight Problems | 42
  Tumor Assessment Week 042: Moderate Problems: number analyzed (Participants) | 145
  Tumor Assessment Week 042: Moderate Problems | 10
  Tumor Assessment Week 042: Severe Problems: number analyzed (Participants) | 145
  Tumor Assessment Week 042: Severe Problems | 3
  Tumor Assessment Week 048: No Problem: number analyzed (Participants) | 126
  Tumor Assessment Week 048: No Problem | 81
  Tumor Assessment Week 048: Slight Problems: number analyzed (Participants) | 126
  Tumor Assessment Week 048: Slight Problems | 34
  Tumor Assessment Week 048: Moderate Problems: number analyzed (Participants) | 126
  Tumor Assessment Week 048: Moderate Problems | 11
  Tumor Assessment Week 054: No Problem: number analyzed (Participants) | 23
  Tumor Assessment Week 054: No Problem | 13
  Tumor Assessment Week 054: Slight Problems: number analyzed (Participants) | 23
  Tumor Assessment Week 054: Slight Problems | 7
  Tumor Assessment Week 054: Moderate Problems: number analyzed (Participants) | 23
  Tumor Assessment Week 054: Moderate Problems | 3
  Tumor Assessment Week 057: No Problem: number analyzed (Participants) | 97
  Tumor Assessment Week 057: No Problem | 68
  Tumor Assessment Week 057: Slight Problems: number analyzed (Participants) | 97
  Tumor Assessment Week 057: Slight Problems | 18
  Tumor Assessment Week 057: Moderate Problems: number analyzed (Participants) | 97
  Tumor Assessment Week 057: Moderate Problems | 9
  Tumor Assessment Week 057: Severe Problems: number analyzed (Participants) | 97
  Tumor Assessment Week 057: Severe Problems | 2
  Tumor Assessment Week 060: No Problem: number analyzed (Participants) | 17
  Tumor Assessment Week 060: No Problem | 13
  Tumor Assessment Week 060: Slight Problems: number analyzed (Participants) | 17
  Tumor Assessment Week 060: Slight Problems | 2
  Tumor Assessment Week 060: Moderate Problems: number analyzed (Participants) | 17
  Tumor Assessment Week 060: Moderate Problems | 2
  Tumor Assessment Week 066: No Problem: number analyzed (Participants) | 88
  Tumor Assessment Week 066: No Problem | 63
  Tumor Assessment Week 066: Slight Problems: number analyzed (Participants) | 88
  Tumor Assessment Week 066: Slight Problems | 15
  Tumor Assessment Week 066: Moderate Problems: number analyzed (Participants) | 88
  Tumor Assessment Week 066: Moderate Problems | 7
  Tumor Assessment Week 066: Severe Problems: number analyzed (Participants) | 88
  Tumor Assessment Week 066: Severe Problems | 2
  Tumor Assessment Week 066: Extreme Problems: number analyzed (Participants) | 88
  Tumor Assessment Week 066: Extreme Problems | 1
  Tumor Assessment Week 072: No Problem: number analyzed (Participants) | 13
  Tumor Assessment Week 072: No Problem | 8
  Tumor Assessment Week 072: Slight Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 072: Slight Problems | 3
  Tumor Assessment Week 072: Moderate Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 072: Moderate Problems | 2
  Tumor Assessment Week 075: No Problem: number analyzed (Participants) | 73
  Tumor Assessment Week 075: No Problem | 51
  Tumor Assessment Week 075: Slight Problems: number analyzed (Participants) | 73
  Tumor Assessment Week 075: Slight Problems | 19
  Tumor Assessment Week 075: Moderate Problems: number analyzed (Participants) | 73
  Tumor Assessment Week 075: Moderate Problems | 1
  Tumor Assessment Week 075: Severe Problems: number analyzed (Participants) | 73
  Tumor Assessment Week 075: Severe Problems | 2
  Tumor Assessment Week 078: No Problem: number analyzed (Participants) | 10
  Tumor Assessment Week 078: No Problem | 7
  Tumor Assessment Week 078: Slight Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 078: Slight Problems | 2
  Tumor Assessment Week 078: Moderate Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 078: Moderate Problems | 1
  Tumor Assessment Week 084: No Problem: number analyzed (Participants) | 67
  Tumor Assessment Week 084: No Problem | 45
  Tumor Assessment Week 084: Slight Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Slight Problems | 14
  Tumor Assessment Week 084: Moderate Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Moderate Problems | 6
  Tumor Assessment Week 084: Severe Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Severe Problems | 1
  Tumor Assessment Week 084: Extreme Problems: number analyzed (Participants) | 67
  Tumor Assessment Week 084: Extreme Problems | 1
  Tumor Assessment Week 090: No Problem: number analyzed (Participants) | 10
  Tumor Assessment Week 090: No Problem | 6
  Tumor Assessment Week 090: Slight Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 090: Slight Problems | 2
  Tumor Assessment Week 090: Moderate Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 090: Moderate Problems | 1
  Tumor Assessment Week 090: Severe Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 090: Severe Problems | 1
  Tumor Assessment Week 093: No Problem: number analyzed (Participants) | 53
  Tumor Assessment Week 093: No Problem | 36
  Tumor Assessment Week 093: Slight Problems: number analyzed (Participants) | 53
  Tumor Assessment Week 093: Slight Problems | 12
  Tumor Assessment Week 093: Moderate Problems: number analyzed (Participants) | 53
  Tumor Assessment Week 093: Moderate Problems | 4
  Tumor Assessment Week 093: Severe Problems: number analyzed (Participants) | 53
  Tumor Assessment Week 093: Severe Problems | 1
  Tumor Assessment Week 096: No Problem: number analyzed (Participants) | 7
  Tumor Assessment Week 096: No Problem | 3
  Tumor Assessment Week 096: Slight Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 096: Slight Problems | 2
  Tumor Assessment Week 096: Moderate Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 096: Moderate Problems | 1
  Tumor Assessment Week 096: Severe Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 096: Severe Problems | 1
  Tumor Assessment Week 102: No Problem: number analyzed (Participants) | 55
  Tumor Assessment Week 102: No Problem | 36
  Tumor Assessment Week 102: Slight Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Slight Problems | 15
  Tumor Assessment Week 102: Moderate Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Moderate Problems | 2
  Tumor Assessment Week 102: Severe Problems: number analyzed (Participants) | 55
  Tumor Assessment Week 102: Severe Problems | 2
  Tumor Assessment Week 108: No Problem: number analyzed (Participants) | 7
  Tumor Assessment Week 108: No Problem | 2
  Tumor Assessment Week 108: Slight Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 108: Slight Problems | 4
  Tumor Assessment Week 108: Severe Problems: number analyzed (Participants) | 7
  Tumor Assessment Week 108: Severe Problems | 1
  Tumor Assessment Week 111: No Problem: number analyzed (Participants) | 40
  Tumor Assessment Week 111: No Problem | 27
  Tumor Assessment Week 111: Slight Problems: number analyzed (Participants) | 40
  Tumor Assessment Week 111: Slight Problems | 9
  Tumor Assessment Week 111: Moderate Problems: number analyzed (Participants) | 40
  Tumor Assessment Week 111: Moderate Problems | 3
  Tumor Assessment Week 111: Severe Problems: number analyzed (Participants) | 41
  Tumor Assessment Week 111: Severe Problems | 1
  Tumor Assessment Week 114: Slight Problems: number analyzed (Participants) | 2
  Tumor Assessment Week 114: Slight Problems | 1
  Tumor Assessment Week 114: Moderate Problems: number analyzed (Participants) | 2
  Tumor Assessment Week 114: Moderate Problems | 1
  Tumor Assessment Week 120: No Problem: number analyzed (Participants) | 38
  Tumor Assessment Week 120: No Problem | 24
  Tumor Assessment Week 120: Slight Problems: number analyzed (Participants) | 38
  Tumor Assessment Week 120: Slight Problems | 11
  Tumor Assessment Week 120: Moderate Problems: number analyzed (Participants) | 38
  Tumor Assessment Week 120: Moderate Problems | 3
  Tumor Assessment Week 126: No Problem: number analyzed (Participants) | 4
  Tumor Assessment Week 126: No Problem | 2
  Tumor Assessment Week 126: Slight Problems: number analyzed (Participants) | 4
  Tumor Assessment Week 126: Slight Problems | 1
  Tumor Assessment Week 126: Moderate Problems: number analyzed (Participants) | 4
  Tumor Assessment Week 126: Moderate Problems | 1
  Tumor Assessment Week 129: No Problem: number analyzed (Participants) | 32
  Tumor Assessment Week 129: No Problem | 21
  Tumor Assessment Week 129: Slight Problems: number analyzed (Participants) | 32
  Tumor Assessment Week 129: Slight Problems | 10
  Tumor Assessment Week 129: Severe Problems: number analyzed (Participants) | 32
  Tumor Assessment Week 129: Severe Problems | 1
  Tumor Assessment Week 132: No Problem: number analyzed (Participants) | 2
  Tumor Assessment Week 132: No Problem | 1
  Tumor Assessment Week 132: Moderate problems: number analyzed (Participants) | 2
  Tumor Assessment Week 132: Moderate problems | 1
  Tumor Assessment Week 138: No Problem: number analyzed (Participants) | 28
  Tumor Assessment Week 138: No Problem | 19
  Tumor Assessment Week 138: Slight Problems: number analyzed (Participants) | 28
  Tumor Assessment Week 138: Slight Problems | 6
  Tumor Assessment Week 138: Moderate Problems: number analyzed (Participants) | 28
  Tumor Assessment Week 138: Moderate Problems | 2
  Tumor Assessment Week 138: Invalid Response: number analyzed (Participants) | 28
  Tumor Assessment Week 138: Invalid Response | 1
  Tumor Assessment Week 144: No Problem: number analyzed (Participants) | 1
  Tumor Assessment Week 144: No Problem | 1
  Tumor Assessment Week 147: No Problem: number analyzed (Participants) | 21
  Tumor Assessment Week 147: No Problem | 14
  Tumor Assessment Week 147: Slight Problems: number analyzed (Participants) | 21
  Tumor Assessment Week 147: Slight Problems | 6
  Tumor Assessment Week 147: Severe Problems: number analyzed (Participants) | 21
  Tumor Assessment Week 147: Severe Problems | 1
  Tumor Assessment Week 156: No Problem: number analyzed (Participants) | 15
  Tumor Assessment Week 156: No Problem | 12
  Tumor Assessment Week 156: Slight Problems: number analyzed (Participants) | 15
  Tumor Assessment Week 156: Slight Problems | 2
  Tumor Assessment Week 156: Moderate Problems: number analyzed (Participants) | 15
  Tumor Assessment Week 156: Moderate Problems | 1
  Tumor Assessment Week 165: No Problem: number analyzed (Participants) | 13
  Tumor Assessment Week 165: No Problem | 8
  Tumor Assessment Week 165: Slight Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Slight Problems | 3
  Tumor Assessment Week 165: Moderate Problems: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Moderate Problems | 1
  Tumor Assessment Week 165: Invalid Response: number analyzed (Participants) | 13
  Tumor Assessment Week 165: Invalid Response | 1
  Tumor Assessment Week 174: No Problem: number analyzed (Participants) | 10
  Tumor Assessment Week 174: No Problem | 8
  Tumor Assessment Week 174: Slight Problems: number analyzed (Participants) | 10
  Tumor Assessment Week 174: Slight Problems | 2
  Tumor Assessment Week 183: No Problem: number analyzed (Participants) | 3
  Tumor Assessment Week 183: No Problem | 2
  Tumor Assessment Week 183: Slight Problems: number analyzed (Participants) | 3
  Tumor Assessment Week 183: Slight Problems | 1

10. Secondary Outcome: EQ-5D-5L Questionnaire - VAS Scores
Description: The EQ-5D-5L was a self-reported health status questionnaire that consisted of six questions used to calculate a health utility score for use in health economic analysis. The EQ-5D-5L has two components: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, as well as a VAS that measures health state. The VAS is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. Values presented after baseline represent the change from baseline.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
score on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 517
  Cycle 2 Day 1 | -0.51 (13.61)
  Tumor Assessment Week 06: number analyzed (Participants) | 425
  Tumor Assessment Week 06 | -1.14 (15.17)
  Tumor Assessment Week 012: number analyzed (Participants) | 309
  Tumor Assessment Week 012 | 0.97 (14.07)
  Tumor Assessment Week 018: number analyzed (Participants) | 251
  Tumor Assessment Week 018 | 2.23 (14.24)
  Tumor Assessment Week 024: number analyzed (Participants) | 212
  Tumor Assessment Week 024 | 1.78 (15.48)
  Tumor Assessment Week 030: number analyzed (Participants) | 179
  Tumor Assessment Week 030 | 3.04 (13.97)
  Tumor Assessment Week 036: number analyzed (Participants) | 157
  Tumor Assessment Week 036 | 2.11 (15.56)
  Tumor Assessment Week 042: number analyzed (Participants) | 141
  Tumor Assessment Week 042 | 3.14 (14.84)
  Tumor Assessment Week 048: number analyzed (Participants) | 125
  Tumor Assessment Week 048 | 2.55 (14.76)
  Tumor Assessment Week 054: number analyzed (Participants) | 22
  Tumor Assessment Week 054 | 0.45 (16.25)
  Tumor Assessment Week 057: number analyzed (Participants) | 95
  Tumor Assessment Week 057 | 4.99 (12.94)
  Tumor Assessment Week 060: number analyzed (Participants) | 17
  Tumor Assessment Week 060 | 6.53 (9.68)
  Tumor Assessment Week 066: number analyzed (Participants) | 85
  Tumor Assessment Week 066 | 2.64 (12.42)
  Tumor Assessment Week 072: number analyzed (Participants) | 13
  Tumor Assessment Week 072 | 2.46 (10.82)
  Tumor Assessment Week 075: number analyzed (Participants) | 71
  Tumor Assessment Week 075 | 3.13 (14.36)
  Tumor Assessment Week 078: number analyzed (Participants) | 10
  Tumor Assessment Week 078 | 6.00 (9.94)
  Tumor Assessment Week 084: number analyzed (Participants) | 66
  Tumor Assessment Week 084 | 4.26 (16.91)
  Tumor Assessment Week 090: number analyzed (Participants) | 10
  Tumor Assessment Week 090 | 2.80 (10.55)
  Tumor Assessment Week 093: number analyzed (Participants) | 51
  Tumor Assessment Week 093 | 5.47 (15.35)
  Tumor Assessment Week 096: number analyzed (Participants) | 7
  Tumor Assessment Week 096 | 6.43 (18.42)
  Tumor Assessment Week 102: number analyzed (Participants) | 53
  Tumor Assessment Week 102 | 4.98 (14.28)
  Tumor Assessment Week 108: number analyzed (Participants) | 7
  Tumor Assessment Week 108 | 10.71 (14.56)
  Tumor Assessment Week 111: number analyzed (Participants) | 39
  Tumor Assessment Week 111 | 4.64 (13.16)
  Tumor Assessment Week 114: number analyzed (Participants) | 2
  Tumor Assessment Week 114 | 15.00 (0.00)
  Tumor Assessment Week 120: number analyzed (Participants) | 37
  Tumor Assessment Week 120 | 5.65 (14.18)
  Tumor Assessment Week 126: number analyzed (Participants) | 4
  Tumor Assessment Week 126 | 16.25 (4.79)
  Tumor Assessment Week 129: number analyzed (Participants) | 31
  Tumor Assessment Week 129 | 4.26 (13.99)
  Tumor Assessment Week 132: number analyzed (Participants) | 2
  Tumor Assessment Week 132 | 12.50 (17.68)
  Tumor Assessment Week 138: number analyzed (Participants) | 27
  Tumor Assessment Week 138 | 2.85 (15.49)
  Tumor Assessment Week 144: number analyzed (Participants) | 1
  Tumor Assessment Week 144 | -8.00 (NA) — Since only 1 participant was analyzed, standard deviation could not be calculated.
  Tumor Assessment Week 147: number analyzed (Participants) | 20
  Tumor Assessment Week 147 | 6.00 (13.14)
  Tumor Assessment Week 156: number analyzed (Participants) | 15
  Tumor Assessment Week 156 | 5.67 (16.24)
  Tumor Assessment Week 165: number analyzed (Participants) | 12
  Tumor Assessment Week 165 | 7.08 (18.52)
  Tumor Assessment Week 174: number analyzed (Participants) | 9
  Tumor Assessment Week 174 | 4.44 (13.33)
  Tumor Assessment Week 183: number analyzed (Participants) | 3
  Tumor Assessment Week 183 | 5.33 (21.57)

11. Secondary Outcome: European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Supplemental Lung Cancer Module (EORTC QLQ-LC13)
Description: The EORTC QLQ-LC13 consisted of 13 items that address key lung cancer symptoms (cough, hemoptysis, dyspnea, and site-specific pain), treatment-related adverse effects (sore mouth, dysphagia, peripheral neuropathy and alopecia) and pain medication. The dysphagia scale is multi-item, while the rest are single-item scales. The scales are linearly transformed so that each score has a range from 0 to 100. A high scale score represents a higher response level (e.g. a high score for global health status represents a high QoL). A high score for the symptom scale represents a high level of symptoms. A >=10-point change in the EORTC scale score was perceived by participants as clinically significant. Values presented after baseline represent the change from baseline.
Time Frame: Day 1 of first 3 cycles (21-day cycle), then every 6 weeks for 48 weeks; thereafter every 9 weeks until disease progression or until treatment discontinuation (up to 4 years)
Population: The safety population was based on all participants who received any dose of atezolizumab during the study treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Units on a scale
  Dyspnoea: Baseline: number analyzed (Participants) | 578
  Dyspnoea: Baseline | 24.82 (21.64)
  Dyspnoea: Cycle (C) 02 Day (D) 01: number analyzed (Participants) | 489
  Dyspnoea: Cycle (C) 02 Day (D) 01 | 2.41 (15.59)
  Dyspnoea: Tumor Assessment Wk 006: number analyzed (Participants) | 329
  Dyspnoea: Tumor Assessment Wk 006 | 1.59 (18.91)
  Dyspnoea: Tumor Assessment Wk 012: number analyzed (Participants) | 216
  Dyspnoea: Tumor Assessment Wk 012 | -0.62 (19.40)
  Dyspnoea: Tumor Assessment Wk 018: number analyzed (Participants) | 178
  Dyspnoea: Tumor Assessment Wk 018 | -0.50 (17.91)
  Dyspnoea: Tumor Assessment Wk 024: number analyzed (Participants) | 145
  Dyspnoea: Tumor Assessment Wk 024 | -2.84 (17.90)
  Dyspnoea: Tumor Assessment Wk 030: number analyzed (Participants) | 114
  Dyspnoea: Tumor Assessment Wk 030 | -1.17 (21.29)
  Dyspnoea: Tumor Assessment Wk 036: number analyzed (Participants) | 91
  Dyspnoea: Tumor Assessment Wk 036 | -3.91 (20.51)
  Dyspnoea: Tumor Assessment Wk 042: number analyzed (Participants) | 84
  Dyspnoea: Tumor Assessment Wk 042 | -3.97 (19.10)
  Dyspnoea: Tumor Assessment Wk 048: number analyzed (Participants) | 70
  Dyspnoea: Tumor Assessment Wk 048 | -3.65 (20.44)
  Dyspnoea: Tumor Assessment Wk 054: number analyzed (Participants) | 14
  Dyspnoea: Tumor Assessment Wk 054 | 2.38 (16.98)
  Dyspnoea: Tumor Assessment Wk 057: number analyzed (Participants) | 55
  Dyspnoea: Tumor Assessment Wk 057 | -5.25 (18.13)
  Dyspnoea: Tumor Assessment Wk 060: number analyzed (Participants) | 10
  Dyspnoea: Tumor Assessment Wk 060 | -1.11 (11.05)
  Dyspnoea: Tumor Assessment Wk 066: number analyzed (Participants) | 51
  Dyspnoea: Tumor Assessment Wk 066 | 1.09 (19.53)
  Dyspnoea: Tumor Assessment Wk 072: number analyzed (Participants) | 7
  Dyspnoea: Tumor Assessment Wk 072 | 4.76 (30.67)
  Dyspnoea: Tumor Assessment Wk 075: number analyzed (Participants) | 40
  Dyspnoea: Tumor Assessment Wk 075 | -2.22 (18.52)
  Dyspnoea: Tumor Assessment Wk 078: number analyzed (Participants) | 5
  Dyspnoea: Tumor Assessment Wk 078 | 0.00 (42.31)
  Dyspnoea: Tumor Assessment Wk 084: number analyzed (Participants) | 38
  Dyspnoea: Tumor Assessment Wk 084 | -2.92 (16.07)
  Dyspnoea: Tumor Assessment Wk 090: number analyzed (Participants) | 5
  Dyspnoea: Tumor Assessment Wk 090 | -17.78 (12.67)
  Dyspnoea: Tumor Assessment Wk 093: number analyzed (Participants) | 28
  Dyspnoea: Tumor Assessment Wk 093 | -3.57 (19.38)
  Dyspnoea: Tumor Assessment Wk 096: number analyzed (Participants) | 5
  Dyspnoea: Tumor Assessment Wk 096 | 13.33 (27.67)
  Dyspnoea: Tumor Assessment Wk 102: number analyzed (Participants) | 28
  Dyspnoea: Tumor Assessment Wk 102 | -5.95 (19.24)
  Dyspnoea: Tumor Assessment Wk 108: number analyzed (Participants) | 5
  Dyspnoea: Tumor Assessment Wk 108 | -8.89 (26.53)
  Dyspnoea: Tumor Assessment Wk 111: number analyzed (Participants) | 21
  Dyspnoea: Tumor Assessment Wk 111 | -6.88 (17.02)
  Dyspnoea: Tumor Assessment Wk 114: number analyzed (Participants) | 2
  Dyspnoea: Tumor Assessment Wk 114 | -16.67 (23.57)
  Dyspnoea: Tumor Assessment Wk 120: number analyzed (Participants) | 19
  Dyspnoea: Tumor Assessment Wk 120 | -5.85 (14.04)
  Dyspnoea: Tumor Assessment Wk 126: number analyzed (Participants) | 3
  Dyspnoea: Tumor Assessment Wk 126 | -18.52 (27.96)
  Dyspnoea: Tumor Assessment Wk 129: number analyzed (Participants) | 17
  Dyspnoea: Tumor Assessment Wk 129 | -7.19 (13.57)
  Dyspnoea: Tumor Assessment Wk 132: number analyzed (Participants) | 1
  Dyspnoea: Tumor Assessment Wk 132 | -22.22
  Dyspnoea: Tumor Assessment Wk 138: number analyzed (Participants) | 13
  Dyspnoea: Tumor Assessment Wk 138 | -1.71 (11.87)
  Dyspnoea: Tumor Assessment Wk 144: number analyzed (Participants) | 1
  Dyspnoea: Tumor Assessment Wk 144 | 0.00
  Dyspnoea: Tumor Assessment Wk 147: number analyzed (Participants) | 9
  Dyspnoea: Tumor Assessment Wk 147 | -3.70 (7.86)
  Dyspnoea: Tumor Assessment Wk 156: number analyzed (Participants) | 8
  Dyspnoea: Tumor Assessment Wk 156 | 6.94 (23.71)
  Dyspnoea: Tumor Assessment Wk 165: number analyzed (Participants) | 3
  Dyspnoea: Tumor Assessment Wk 165 | 3.70 (23.13)
  Dyspnoea: Tumor Assessment Wk 174: number analyzed (Participants) | 1
  Dyspnoea: Tumor Assessment Wk 174 | 0.00
  Dyspnoea: Tumor Assessment Wk 183: number analyzed (Participants) | 1
  Dyspnoea: Tumor Assessment Wk 183 | -11.11
  Coughing: Baseline: number analyzed (Participants) | 587
  Coughing: Baseline | 33.84 (25.94)
  Coughing: C2D1: number analyzed (Participants) | 501
  Coughing: C2D1 | 0.80 (21.89)
  Coughing: Tumor Assessment Wk 006: number analyzed (Participants) | 341
  Coughing: Tumor Assessment Wk 006 | -0.68 (24.84)
  Coughing: Tumor Assessment Wk 012: number analyzed (Participants) | 225
  Coughing: Tumor Assessment Wk 012 | -4.44 (28.35)
  Coughing: Tumor Assessment Wk 018: number analyzed (Participants) | 182
  Coughing: Tumor Assessment Wk 018 | -7.88 (25.61)
  Coughing: Tumor Assessment Wk 024: number analyzed (Participants) | 149
  Coughing: Tumor Assessment Wk 024 | -7.83 (26.95)
  Coughing: Tumor Assessment Wk 030: number analyzed (Participants) | 116
  Coughing: Tumor Assessment Wk 030 | -7.18 (26.30)
  Coughing: Tumor Assessment Wk 036: number analyzed (Participants) | 93
  Coughing: Tumor Assessment Wk 036 | -9.32 (25.71)
  Coughing: Tumor Assessment Wk 042: number analyzed (Participants) | 86
  Coughing: Tumor Assessment Wk 042 | -13.18 (25.71)
  Coughing: Tumor Assessment Wk 048: number analyzed (Participants) | 72
  Coughing: Tumor Assessment Wk 048 | -9.26 (30.76)
  Coughing: Tumor Assessment Wk 054: number analyzed (Participants) | 14
  Coughing: Tumor Assessment Wk 054 | -2.38 (24.33)
  Coughing: Tumor Assessment Wk 057: number analyzed (Participants) | 58
  Coughing: Tumor Assessment Wk 057 | -13.22 (28.57)
  Coughing: Tumor Assessment Wk 060: number analyzed (Participants) | 11
  Coughing: Tumor Assessment Wk 060 | -9.09 (21.56)
  Coughing: Tumor Assessment Wk 066: number analyzed (Participants) | 53
  Coughing: Tumor Assessment Wk 066 | -10.69 (28.32)
  Coughing: Tumor Assessment Wk 072: number analyzed (Participants) | 7
  Coughing: Tumor Assessment Wk 072 | -4.76 (23.00)
  Coughing: Tumor Assessment Wk 075: number analyzed (Participants) | 40
  Coughing: Tumor Assessment Wk 075 | -18.33 (28.19)
  Coughing: Tumor Assessment Wk 078: number analyzed (Participants) | 5
  Coughing: Tumor Assessment Wk 078 | 0.00 (33.33)
  Coughing: Tumor Assessment Wk 084: number analyzed (Participants) | 38
  Coughing: Tumor Assessment Wk 084 | -16.67 (31.72)
  Coughing: Tumor Assessment Wk 090: number analyzed (Participants) | 6
  Coughing: Tumor Assessment Wk 090 | -16.67 (18.26)
  Coughing: Tumor Assessment Wk 093: number analyzed (Participants) | 28
  Coughing: Tumor Assessment Wk 093 | -16.67 (30.77)
  Coughing: Tumor Assessment Wk 096: number analyzed (Participants) | 5
  Coughing: Tumor Assessment Wk 096 | 6.67 (14.91)
  Coughing: Tumor Assessment Wk 102: number analyzed (Participants) | 28
  Coughing: Tumor Assessment Wk 102 | -23.81 (25.43)
  Coughing: Tumor Assessment Wk 108: number analyzed (Participants) | 5
  Coughing: Tumor Assessment Wk 108 | -6.67 (27.89)
  Coughing: Tumor Assessment Wk 111: number analyzed (Participants) | 21
  Coughing: Tumor Assessment Wk 111 | -11.11 (30.43)
  Coughing: Tumor Assessment Wk 114: number analyzed (Participants) | 2
  Coughing: Tumor Assessment Wk 114 | -16.67 (23.57)
  Coughing: Tumor Assessment Wk 120: number analyzed (Participants) | 19
  Coughing: Tumor Assessment Wk 120 | -12.28 (29.84)
  Coughing: Tumor Assessment Wk 126: number analyzed (Participants) | 3
  Coughing: Tumor Assessment Wk 126 | 0.00 (33.33)
  Coughing: Tumor Assessment Wk 129: number analyzed (Participants) | 17
  Coughing: Tumor Assessment Wk 129 | -11.76 (26.20)
  Coughing: Tumor Assessment Wk 132: number analyzed (Participants) | 1
  Coughing: Tumor Assessment Wk 132 | 0.00
  Coughing: Tumor Assessment Wk 138: number analyzed (Participants) | 14
  Coughing: Tumor Assessment Wk 138 | -14.29 (31.25)
  Coughing: Tumor Assessment Wk 144: number analyzed (Participants) | 1
  Coughing: Tumor Assessment Wk 144 | 33.33
  Coughing: Tumor Assessment Wk 147: number analyzed (Participants) | 9
  Coughing: Tumor Assessment Wk 147 | -22.22 (40.82)
  Coughing: Tumor Assessment Wk 156: number analyzed (Participants) | 8
  Coughing: Tumor Assessment Wk 156 | -12.50 (53.27)
  Coughing: Tumor Assessment Wk 165: number analyzed (Participants) | 3
  Coughing: Tumor Assessment Wk 165 | 0.00 (33.33)
  Coughing: Tumor Assessment Wk 174: number analyzed (Participants) | 1
  Coughing: Tumor Assessment Wk 174 | 33.33
  Coughing: Tumor Assessment Wk 183: number analyzed (Participants) | 1
  Coughing: Tumor Assessment Wk 183 | 0.00
  Haemoptysis: Baseline: number analyzed (Participants) | 585
  Haemoptysis: Baseline | 3.02 (10.15)
  Haemoptysis: C2D1: number analyzed (Participants) | 501
  Haemoptysis: C2D1 | 0.60 (9.05)
  Haemoptysis: Tumor Assessment Wk 006: number analyzed (Participants) | 336
  Haemoptysis: Tumor Assessment Wk 006 | 0.10 (9.81)
  Haemoptysis: Tumor Assessment Wk 012: number analyzed (Participants) | 222
  Haemoptysis: Tumor Assessment Wk 012 | 0.15 (9.77)
  Haemoptysis: Tumor Assessment Wk 018: number analyzed (Participants) | 181
  Haemoptysis: Tumor Assessment Wk 018 | -0.18 (8.96)
  Haemoptysis: Tumor Assessment Wk 024: number analyzed (Participants) | 149
  Haemoptysis: Tumor Assessment Wk 024 | -0.67 (9.06)
  Haemoptysis: Tumor Assessment Wk 030: number analyzed (Participants) | 116
  Haemoptysis: Tumor Assessment Wk 030 | -0.29 (10.31)
  Haemoptysis: Tumor Assessment Wk 036: number analyzed (Participants) | 93
  Haemoptysis: Tumor Assessment Wk 036 | -1.79 (10.27)
  Haemoptysis: Tumor Assessment Wk 042: number analyzed (Participants) | 86
  Haemoptysis: Tumor Assessment Wk 042 | 0.00 (11.43)
  Haemoptysis: Tumor Assessment Wk 048: number analyzed (Participants) | 72
  Haemoptysis: Tumor Assessment Wk 048 | -0.46 (8.83)
  Haemoptysis: Tumor Assessment Wk 054: number analyzed (Participants) | 14
  Haemoptysis: Tumor Assessment Wk 054 | 0.00 (13.07)
  Haemoptysis: Tumor Assessment Wk 057: number analyzed (Participants) | 57
  Haemoptysis: Tumor Assessment Wk 057 | 0.00 (10.91)
  Haemoptysis: Tumor Assessment Wk 060: number analyzed (Participants) | 11
  Haemoptysis: Tumor Assessment Wk 060 | 0.00 (14.91)
  Haemoptysis: Tumor Assessment Wk 066: number analyzed (Participants) | 53
  Haemoptysis: Tumor Assessment Wk 066 | -2.52 (8.89)
  Haemoptysis: Tumor Assessment Wk 072: number analyzed (Participants) | 7
  Haemoptysis: Tumor Assessment Wk 072 | 0.00 (0.00)
  Haemoptysis: Tumor Assessment Wk 075: number analyzed (Participants) | 40
  Haemoptysis: Tumor Assessment Wk 075 | -3.33 (10.13)
  Haemoptysis: Tumor Assessment Wk 078: number analyzed (Participants) | 5
  Haemoptysis: Tumor Assessment Wk 078 | 0.00 (0.00)
  Haemoptysis: Tumor Assessment Wk 084: number analyzed (Participants) | 38
  Haemoptysis: Tumor Assessment Wk 084 | -2.63 (9.11)
  Haemoptysis: Tumor Assessment Wk 090: number analyzed (Participants) | 6
  Haemoptysis: Tumor Assessment Wk 090 | 5.56 (13.61)
  Haemoptysis: Tumor Assessment Wk 093: number analyzed (Participants) | 28
  Haemoptysis: Tumor Assessment Wk 093 | 1.19 (14.29)
  Haemoptysis: Tumor Assessment Wk 096: number analyzed (Participants) | 5
  Haemoptysis: Tumor Assessment Wk 096 | 0.00 (0.00)
  Haemoptysis: Tumor Assessment Wk 102: number analyzed (Participants) | 28
  Haemoptysis: Tumor Assessment Wk 102 | -2.38 (8.74)
  Haemoptysis: Tumor Assessment Wk 108: number analyzed (Participants) | 5
  Haemoptysis: Tumor Assessment Wk 108 | 0.00 (0.00)
  Haemoptysis: Tumor Assessment Wk 111: number analyzed (Participants) | 21
  Haemoptysis: Tumor Assessment Wk 111 | -3.17 (10.03)
  Haemoptysis: Tumor Assessment Wk 114: number analyzed (Participants) | 2
  Haemoptysis: Tumor Assessment Wk 114 | 0.00 (0.00)
  Haemoptysis: Tumor Assessment Wk 120: number analyzed (Participants) | 19
  Haemoptysis: Tumor Assessment Wk 120 | -1.75 (13.49)
  Haemoptysis: Tumor Assessment Wk 126: number analyzed (Participants) | 3
  Haemoptysis: Tumor Assessment Wk 126 | 0.00 (0.00)
  Haemoptysis: Tumor Assessment Wk 129: number analyzed (Participants) | 17
  Haemoptysis: Tumor Assessment Wk 129 | -1.96 (14.29)
  Haemoptysis: Tumor Assessment Wk 132: number analyzed (Participants) | 1
  Haemoptysis: Tumor Assessment Wk 132 | 0.00
  Haemoptysis: Tumor Assessment Wk 138: number analyzed (Participants) | 14
  Haemoptysis: Tumor Assessment Wk 138 | -2.38 (15.82)
  Haemoptysis: Tumor Assessment Wk 144: number analyzed (Participants) | 1
  Haemoptysis: Tumor Assessment Wk 144 | 0.00
  Haemoptysis: Tumor Assessment Wk 147: number analyzed (Participants) | 9
  Haemoptysis: Tumor Assessment Wk 147 | 0.00 (16.67)
  Haemoptysis: Tumor Assessment Wk 156: number analyzed (Participants) | 8
  Haemoptysis: Tumor Assessment Wk 156 | 0.00 (0.00)
  Haemoptysis: Tumor Assessment Wk 165: number analyzed (Participants) | 3
  Haemoptysis: Tumor Assessment Wk 165 | 0.00 (33.33)
  Haemoptysis: Tumor Assessment Wk 174: number analyzed (Participants) | 1
  Haemoptysis: Tumor Assessment Wk 174 | -33.33
  Haemoptysis: Tumor Assessment Wk 183: number analyzed (Participants) | 1
  Haemoptysis: Tumor Assessment Wk 183 | 0.00
  Sore mouth: Baseline: number analyzed (Participants) | 587
  Sore mouth: Baseline | 3.58 (12.33)
  Sore mouth: C2D1: number analyzed (Participants) | 501
  Sore mouth: C2D1 | 0.67 (15.76)
  Sore mouth: Tumor Assessment Wk 006: number analyzed (Participants) | 337
  Sore mouth: Tumor Assessment Wk 006 | 0.49 (16.95)
  Sore mouth: Tumor Assessment Wk 012: number analyzed (Participants) | 220
  Sore mouth: Tumor Assessment Wk 012 | 0.00 (16.55)
  Sore mouth: Tumor Assessment Wk 018: number analyzed (Participants) | 182
  Sore mouth: Tumor Assessment Wk 018 | -0.73 (14.00)
  Sore mouth: Tumor Assessment Wk 024: number analyzed (Participants) | 148
  Sore mouth: Tumor Assessment Wk 024 | -1.13 (14.24)
  Sore mouth: Tumor Assessment Wk 030: number analyzed (Participants) | 115
  Sore mouth: Tumor Assessment Wk 030 | -2.03 (14.16)
  Sore mouth: Tumor Assessment Wk 036: number analyzed (Participants) | 92
  Sore mouth: Tumor Assessment Wk 036 | -2.54 (15.02)
  Sore mouth: Tumor Assessment Wk 042: number analyzed (Participants) | 85
  Sore mouth: Tumor Assessment Wk 042 | -1.57 (16.99)
  Sore mouth: Tumor Assessment Wk 048: number analyzed (Participants) | 70
  Sore mouth: Tumor Assessment Wk 048 | -4.29 (15.97)
  Sore mouth: Tumor Assessment Wk 054: number analyzed (Participants) | 13
  Sore mouth: Tumor Assessment Wk 054 | 2.56 (16.45)
  Sore mouth: Tumor Assessment Wk 057: number analyzed (Participants) | 57
  Sore mouth: Tumor Assessment Wk 057 | -1.75 (11.65)
  Sore mouth: Tumor Assessment Wk 060: number analyzed (Participants) | 10
  Sore mouth: Tumor Assessment Wk 060 | -3.33 (10.54)
  Sore mouth: Tumor Assessment Wk 066: number analyzed (Participants) | 52
  Sore mouth: Tumor Assessment Wk 066 | -2.56 (14.53)
  Sore mouth: Tumor Assessment Wk 072: number analyzed (Participants) | 7
  Sore mouth: Tumor Assessment Wk 072 | 0.00 (0.00)
  Sore mouth: Tumor Assessment Wk 075: number analyzed (Participants) | 40
  Sore mouth: Tumor Assessment Wk 075 | -2.50 (13.89)
  Sore mouth: Tumor Assessment Wk 078: number analyzed (Participants) | 5
  Sore mouth: Tumor Assessment Wk 078 | 6.67 (14.91)
  Sore mouth: Tumor Assessment Wk 084: number analyzed (Participants) | 38
  Sore mouth: Tumor Assessment Wk 084 | -1.75 (13.30)
  Sore mouth: Tumor Assessment Wk 090: number analyzed (Participants) | 6
  Sore mouth: Tumor Assessment Wk 090 | 0.00 (0.00)
  Sore mouth: Tumor Assessment Wk 093: number analyzed (Participants) | 28
  Sore mouth: Tumor Assessment Wk 093 | 2.38 (8.74)
  Sore mouth: Tumor Assessment Wk 096: number analyzed (Participants) | 5
  Sore mouth: Tumor Assessment Wk 096 | 0.00 (0.00)
  Sore mouth: Tumor Assessment Wk 102: number analyzed (Participants) | 28
  Sore mouth: Tumor Assessment Wk 102 | 1.19 (6.30)
  Sore mouth: Tumor Assessment Wk 108: number analyzed (Participants) | 5
  Sore mouth: Tumor Assessment Wk 108 | 0.00 (0.00)
  Sore mouth: Tumor Assessment Wk 111: number analyzed (Participants) | 21
  Sore mouth: Tumor Assessment Wk 111 | 3.17 (10.03)
  Sore mouth: Tumor Assessment Wk 114: number analyzed (Participants) | 2
  Sore mouth: Tumor Assessment Wk 114 | 33.33 (47.14)
  Sore mouth: Tumor Assessment Wk 120: number analyzed (Participants) | 19
  Sore mouth: Tumor Assessment Wk 120 | 7.02 (17.84)
  Sore mouth: Tumor Assessment Wk 126: number analyzed (Participants) | 3
  Sore mouth: Tumor Assessment Wk 126 | 11.11 (19.25)
  Sore mouth: Tumor Assessment Wk 129: number analyzed (Participants) | 17
  Sore mouth: Tumor Assessment Wk 129 | 0.00 (0.00)
  Sore mouth: Tumor Assessment Wk 132: number analyzed (Participants) | 1
  Sore mouth: Tumor Assessment Wk 132 | 33.33
  Sore mouth: Tumor Assessment Wk 138: number analyzed (Participants) | 14
  Sore mouth: Tumor Assessment Wk 138 | 2.38 (8.91)
  Sore mouth: Tumor Assessment Wk 144: number analyzed (Participants) | 1
  Sore mouth: Tumor Assessment Wk 144 | 0.00
  Sore mouth: Tumor Assessment Wk 147: number analyzed (Participants) | 9
  Sore mouth: Tumor Assessment Wk 147 | 0.00 (0.00)
  Sore mouth: Tumor Assessment Wk 156: number analyzed (Participants) | 8
  Sore mouth: Tumor Assessment Wk 156 | 0.00 (0.00)
  Sore mouth: Tumor Assessment Wk 165: number analyzed (Participants) | 3
  Sore mouth: Tumor Assessment Wk 165 | 0.00 (0.00)
  Sore mouth: Tumor Assessment Wk 174: number analyzed (Participants) | 1
  Sore mouth: Tumor Assessment Wk 174 | 0.00
  Sore mouth: Tumor Assessment Wk 183: number analyzed (Participants) | 1
  Sore mouth: Tumor Assessment Wk 183 | 0.00
  Dysphagia: Baseline: number analyzed (Participants) | 586
  Dysphagia: Baseline | 5.46 (14.73)
  Dysphagia: C2D1: number analyzed (Participants) | 500
  Dysphagia: C2D1 | 0.20 (13.92)
  Dysphagia: Tumor Assessment Wk 006: number analyzed (Participants) | 339
  Dysphagia: Tumor Assessment Wk 006 | -1.38 (13.74)
  Dysphagia: Tumor Assessment Wk 012: number analyzed (Participants) | 222
  Dysphagia: Tumor Assessment Wk 012 | -0.15 (16.63)
  Dysphagia: Tumor Assessment Wk 018: number analyzed (Participants) | 181
  Dysphagia: Tumor Assessment Wk 018 | 0.74 (16.08)
  Dysphagia: Tumor Assessment Wk 024: number analyzed (Participants) | 147
  Dysphagia: Tumor Assessment Wk 024 | -1.59 (11.26)
  Dysphagia: Tumor Assessment Wk 030: number analyzed (Participants) | 114
  Dysphagia: Tumor Assessment Wk 030 | -1.46 (10.30)
  Dysphagia: Tumor Assessment Wk 036: number analyzed (Participants) | 91
  Dysphagia: Tumor Assessment Wk 036 | -1.83 (16.00)
  Dysphagia: Tumor Assessment Wk 042: number analyzed (Participants) | 84
  Dysphagia: Tumor Assessment Wk 042 | -1.59 (13.60)
  Dysphagia: Tumor Assessment Wk 048: number analyzed (Participants) | 70
  Dysphagia: Tumor Assessment Wk 048 | -0.48 (15.53)
  Dysphagia: Tumor Assessment Wk 054: number analyzed (Participants) | 13
  Dysphagia: Tumor Assessment Wk 054 | -2.56 (9.25)
  Dysphagia: Tumor Assessment Wk 057: number analyzed (Participants) | 57
  Dysphagia: Tumor Assessment Wk 057 | -0.58 (9.94)
  Dysphagia: Tumor Assessment Wk 060: number analyzed (Participants) | 10
  Dysphagia: Tumor Assessment Wk 060 | 0.00 (0.00)
  Dysphagia: Tumor Assessment Wk 066: number analyzed (Participants) | 52
  Dysphagia: Tumor Assessment Wk 066 | -1.28 (11.36)
  Dysphagia: Tumor Assessment Wk 072: number analyzed (Participants) | 7
  Dysphagia: Tumor Assessment Wk 072 | 0.00 (0.00)
  Dysphagia: Tumor Assessment Wk 075: number analyzed (Participants) | 40
  Dysphagia: Tumor Assessment Wk 075 | 0.00 (15.10)
  Dysphagia: Tumor Assessment Wk 078: number analyzed (Participants) | 4
  Dysphagia: Tumor Assessment Wk 078 | 0.00 (0.00)
  Dysphagia: Tumor Assessment Wk 084: number analyzed (Participants) | 38
  Dysphagia: Tumor Assessment Wk 084 | -2.63 (11.96)
  Dysphagia: Tumor Assessment Wk 090: number analyzed (Participants) | 6
  Dysphagia: Tumor Assessment Wk 090 | 0.00 (0.00)
  Dysphagia: Tumor Assessment Wk 093: number analyzed (Participants) | 28
  Dysphagia: Tumor Assessment Wk 093 | -2.38 (8.74)
  Dysphagia: Tumor Assessment Wk 096: number analyzed (Participants) | 5
  Dysphagia: Tumor Assessment Wk 096 | 6.67 (14.91)
  Dysphagia: Tumor Assessment Wk 102: number analyzed (Participants) | 28
  Dysphagia: Tumor Assessment Wk 102 | -2.38 (8.74)
  Dysphagia: Tumor Assessment Wk 108: number analyzed (Participants) | 5
  Dysphagia: Tumor Assessment Wk 108 | 0.00 (0.00)
  Dysphagia: Tumor Assessment Wk 111: number analyzed (Participants) | 21
  Dysphagia: Tumor Assessment Wk 111 | 0.00 (10.54)
  Dysphagia: Tumor Assessment Wk 114: number analyzed (Participants) | 2
  Dysphagia: Tumor Assessment Wk 114 | 0.00 (0.00)
  Dysphagia: Tumor Assessment Wk 120: number analyzed (Participants) | 19
  Dysphagia: Tumor Assessment Wk 120 | -1.75 (7.65)
  Dysphagia: Tumor Assessment Wk 126: number analyzed (Participants) | 3
  Dysphagia: Tumor Assessment Wk 126 | 0.00 (0.00)
  Dysphagia: Tumor Assessment Wk 129: number analyzed (Participants) | 17
  Dysphagia: Tumor Assessment Wk 129 | 0.00 (0.00)
  Dysphagia: Tumor Assessment Wk 132: number analyzed (Participants) | 1
  Dysphagia: Tumor Assessment Wk 132 | 0.00
  Dysphagia: Tumor Assessment Wk 138: number analyzed (Participants) | 14
  Dysphagia: Tumor Assessment Wk 138 | 0.00 (0.00)
  Dysphagia: Tumor Assessment Wk 144: number analyzed (Participants) | 1
  Dysphagia: Tumor Assessment Wk 144 | 0.00
  Dysphagia: Tumor Assessment Wk 147: number analyzed (Participants) | 9
  Dysphagia: Tumor Assessment Wk 147 | 0.00 (0.00)
  Dysphagia: Tumor Assessment Wk 156: number analyzed (Participants) | 8
  Dysphagia: Tumor Assessment Wk 156 | 4.17 (11.79)
  Dysphagia: Tumor Assessment Wk 165: number analyzed (Participants) | 3
  Dysphagia: Tumor Assessment Wk 165 | 0.00 (0.00)
  Dysphagia: Tumor Assessment Wk 174: number analyzed (Participants) | 1
  Dysphagia: Tumor Assessment Wk 174 | 0.00
  Dysphagia: Tumor Assessment Wk 183: number analyzed (Participants) | 1
  Dysphagia: Tumor Assessment Wk 183 | 0.00
  Peripheral neuropathy: Baseline: number analyzed (Participants) | 589
  Peripheral neuropathy: Baseline | 17.77 (26.96)
  Peripheral neuropathy: C2D1: number analyzed (Participants) | 504
  Peripheral neuropathy: C2D1 | -0.20 (22.29)
  Peripheral neuropathy: Tumor Assessment Wk 006: number analyzed (Participants) | 342
  Peripheral neuropathy: Tumor Assessment Wk 006 | -0.58 (21.80)
  Peripheral neuropathy: Tumor Assessment Wk 012: number analyzed (Participants) | 223
  Peripheral neuropathy: Tumor Assessment Wk 012 | 0.15 (24.20)
  Peripheral neuropathy: Tumor Assessment Wk 018: number analyzed (Participants) | 182
  Peripheral neuropathy: Tumor Assessment Wk 018 | -2.56 (26.56)
  Peripheral neuropathy: Tumor Assessment Wk 024: number analyzed (Participants) | 148
  Peripheral neuropathy: Tumor Assessment Wk 024 | -3.15 (25.30)
  Peripheral neuropathy: Tumor Assessment Wk 030: number analyzed (Participants) | 115
  Peripheral neuropathy: Tumor Assessment Wk 030 | -3.19 (24.17)
  Peripheral neuropathy: Tumor Assessment Wk 036: number analyzed (Participants) | 91
  Peripheral neuropathy: Tumor Assessment Wk 036 | -6.23 (25.29)
  Peripheral neuropathy: Tumor Assessment Wk 042: number analyzed (Participants) | 85
  Peripheral neuropathy: Tumor Assessment Wk 042 | -7.45 (28.35)
  Peripheral neuropathy: Tumor Assessment Wk 048: number analyzed (Participants) | 71
  Peripheral neuropathy: Tumor Assessment Wk 048 | -8.92 (27.58)
  Peripheral neuropathy: Tumor Assessment Wk 054: number analyzed (Participants) | 13
  Peripheral neuropathy: Tumor Assessment Wk 054 | -7.69 (19.97)
  Peripheral neuropathy: Tumor Assessment Wk 057: number analyzed (Participants) | 58
  Peripheral neuropathy: Tumor Assessment Wk 057 | -6.32 (20.19)
  Peripheral neuropathy: Tumor Assessment Wk 060: number analyzed (Participants) | 10
  Peripheral neuropathy: Tumor Assessment Wk 060 | -13.33 (17.21)
  Peripheral neuropathy: Tumor Assessment Wk 066: number analyzed (Participants) | 52
  Peripheral neuropathy: Tumor Assessment Wk 066 | -3.85 (22.53)
  Peripheral neuropathy: Tumor Assessment Wk 072: number analyzed (Participants) | 7
  Peripheral neuropathy: Tumor Assessment Wk 072 | -4.76 (23.00)
  Peripheral neuropathy: Tumor Assessment Wk 075: number analyzed (Participants) | 40
  Peripheral neuropathy: Tumor Assessment Wk 075 | -10.83 (26.57)
  Peripheral neuropathy: Tumor Assessment Wk 078: number analyzed (Participants) | 5
  Peripheral neuropathy: Tumor Assessment Wk 078 | -6.67 (27.89)
  Peripheral neuropathy: Tumor Assessment Wk 084: number analyzed (Participants) | 38
  Peripheral neuropathy: Tumor Assessment Wk 084 | -9.65 (28.90)
  Peripheral neuropathy: Tumor Assessment Wk 090: number analyzed (Participants) | 6
  Peripheral neuropathy: Tumor Assessment Wk 090 | 0.00 (21.08)
  Peripheral neuropathy: Tumor Assessment Wk 093: number analyzed (Participants) | 28
  Peripheral neuropathy: Tumor Assessment Wk 093 | -5.95 (30.16)
  Peripheral neuropathy: Tumor Assessment Wk 096: number analyzed (Participants) | 5
  Peripheral neuropathy: Tumor Assessment Wk 096 | 6.67 (14.91)
  Peripheral neuropathy: Tumor Assessment Wk 102: number analyzed (Participants) | 28
  Peripheral neuropathy: Tumor Assessment Wk 102 | -8.33 (26.64)
  Peripheral neuropathy: Tumor Assessment Wk 108: number analyzed (Participants) | 5
  Peripheral neuropathy: Tumor Assessment Wk 108 | -6.67 (14.91)
  Peripheral neuropathy: Tumor Assessment Wk 111: number analyzed (Participants) | 21
  Peripheral neuropathy: Tumor Assessment Wk 111 | -14.29 (34.27)
  Peripheral neuropathy: Tumor Assessment Wk 114: number analyzed (Participants) | 2
  Peripheral neuropathy: Tumor Assessment Wk 114 | -16.67 (23.57)
  Peripheral neuropathy: Tumor Assessment Wk 120: number analyzed (Participants) | 19
  Peripheral neuropathy: Tumor Assessment Wk 120 | -14.04 (32.04)
  Peripheral neuropathy: Tumor Assessment Wk 126: number analyzed (Participants) | 3
  Peripheral neuropathy: Tumor Assessment Wk 126 | -11.11 (19.25)
  Peripheral neuropathy: Tumor Assessment Wk 129: number analyzed (Participants) | 17
  Peripheral neuropathy: Tumor Assessment Wk 129 | -7.84 (25.08)
  Peripheral neuropathy: Tumor Assessment Wk 132: number analyzed (Participants) | 1
  Peripheral neuropathy: Tumor Assessment Wk 132 | 0.00
  Peripheral neuropathy: Tumor Assessment Wk 138: number analyzed (Participants) | 14
  Peripheral neuropathy: Tumor Assessment Wk 138 | -19.05 (33.88)
  Peripheral neuropathy: Tumor Assessment Wk 144: number analyzed (Participants) | 1
  Peripheral neuropathy: Tumor Assessment Wk 144 | 0.00
  Peripheral neuropathy: Tumor Assessment Wk 147: number analyzed (Participants) | 9
  Peripheral neuropathy: Tumor Assessment Wk 147 | -22.22 (40.82)
  Peripheral neuropathy: Tumor Assessment Wk 156: number analyzed (Participants) | 8
  Peripheral neuropathy: Tumor Assessment Wk 156 | -12.50 (50.20)
  Peripheral neuropathy: Tumor Assessment Wk 165: number analyzed (Participants) | 3
  Peripheral neuropathy: Tumor Assessment Wk 165 | 11.11 (19.25)
  Peripheral neuropathy: Tumor Assessment Wk 174: number analyzed (Participants) | 1
  Peripheral neuropathy: Tumor Assessment Wk 174 | 33.33
  Peripheral neuropathy: Tumor Assessment Wk 183: number analyzed (Participants) | 1
  Peripheral neuropathy: Tumor Assessment Wk 183 | 33.33
  Alopecia: Baseline: number analyzed (Participants) | 588
  Alopecia: Baseline | 13.95 (27.14)
  Alopecia: C2D1: number analyzed (Participants) | 502
  Alopecia: C2D1 | -5.64 (24.32)
  Alopecia: Tumor Assessment Wk 006: number analyzed (Participants) | 340
  Alopecia: Tumor Assessment Wk 006 | -4.31 (24.84)
  Alopecia: Tumor Assessment Wk 012: number analyzed (Participants) | 223
  Alopecia: Tumor Assessment Wk 012 | -5.98 (25.39)
  Alopecia: Tumor Assessment Wk 018: number analyzed (Participants) | 180
  Alopecia: Tumor Assessment Wk 018 | -6.85 (24.59)
  Alopecia: Tumor Assessment Wk 024: number analyzed (Participants) | 148
  Alopecia: Tumor Assessment Wk 024 | -8.11 (24.16)
  Alopecia: Tumor Assessment Wk 030: number analyzed (Participants) | 115
  Alopecia: Tumor Assessment Wk 030 | -6.96 (25.93)
  Alopecia: Tumor Assessment Wk 036: number analyzed (Participants) | 92
  Alopecia: Tumor Assessment Wk 036 | -6.52 (25.79)
  Alopecia: Tumor Assessment Wk 042: number analyzed (Participants) | 85
  Alopecia: Tumor Assessment Wk 042 | -6.67 (26.13)
  Alopecia: Tumor Assessment Wk 048: number analyzed (Participants) | 71
  Alopecia: Tumor Assessment Wk 048 | -7.51 (26.55)
  Alopecia: Tumor Assessment Wk 054: number analyzed (Participants) | 13
  Alopecia: Tumor Assessment Wk 054 | 2.56 (9.25)
  Alopecia: Tumor Assessment Wk 057: number analyzed (Participants) | 57
  Alopecia: Tumor Assessment Wk 057 | -6.43 (27.77)
  Alopecia: Tumor Assessment Wk 060: number analyzed (Participants) | 10
  Alopecia: Tumor Assessment Wk 060 | 0.00 (15.71)
  Alopecia: Tumor Assessment Wk 066: number analyzed (Participants) | 52
  Alopecia: Tumor Assessment Wk 066 | -6.41 (26.44)
  Alopecia: Tumor Assessment Wk 072: number analyzed (Participants) | 7
  Alopecia: Tumor Assessment Wk 072 | 9.52 (16.27)
  Alopecia: Tumor Assessment Wk 075: number analyzed (Participants) | 40
  Alopecia: Tumor Assessment Wk 075 | -6.67 (27.43)
  Alopecia: Tumor Assessment Wk 078: number analyzed (Participants) | 5
  Alopecia: Tumor Assessment Wk 078 | 13.33 (18.26)
  Alopecia: Tumor Assessment Wk 084: number analyzed (Participants) | 38
  Alopecia: Tumor Assessment Wk 084 | -6.14 (26.68)
  Alopecia: Tumor Assessment Wk 090: number analyzed (Participants) | 6
  Alopecia: Tumor Assessment Wk 090 | 5.56 (13.61)
  Alopecia: Tumor Assessment Wk 093: number analyzed (Participants) | 28
  Alopecia: Tumor Assessment Wk 093 | -4.76 (28.28)
  Alopecia: Tumor Assessment Wk 096: number analyzed (Participants) | 5
  Alopecia: Tumor Assessment Wk 096 | 6.67 (14.91)
  Alopecia: Tumor Assessment Wk 102: number analyzed (Participants) | 28
  Alopecia: Tumor Assessment Wk 102 | -4.76 (26.78)
  Alopecia: Tumor Assessment Wk 108: number analyzed (Participants) | 5
  Alopecia: Tumor Assessment Wk 108 | 20.00 (18.26)
  Alopecia: Tumor Assessment Wk 111: number analyzed (Participants) | 21
  Alopecia: Tumor Assessment Wk 111 | -3.17 (27.70)
  Alopecia: Tumor Assessment Wk 114: number analyzed (Participants) | 2
  Alopecia: Tumor Assessment Wk 114 | 16.67 (23.57)
  Alopecia: Tumor Assessment Wk 120: number analyzed (Participants) | 19
  Alopecia: Tumor Assessment Wk 120 | 3.51 (29.18)
  Alopecia: Tumor Assessment Wk 126: number analyzed (Participants) | 3
  Alopecia: Tumor Assessment Wk 126 | 22.22 (19.25)
  Alopecia: Tumor Assessment Wk 129: number analyzed (Participants) | 17
  Alopecia: Tumor Assessment Wk 129 | 5.88 (17.62)
  Alopecia: Tumor Assessment Wk 132: number analyzed (Participants) | 1
  Alopecia: Tumor Assessment Wk 132 | 0.00
  Alopecia: Tumor Assessment Wk 138: number analyzed (Participants) | 14
  Alopecia: Tumor Assessment Wk 138 | -4.76 (28.81)
  Alopecia: Tumor Assessment Wk 144: number analyzed (Participants) | 1
  Alopecia: Tumor Assessment Wk 144 | 0.00
  Alopecia: Tumor Assessment Wk 147: number analyzed (Participants) | 9
  Alopecia: Tumor Assessment Wk 147 | -7.41 (36.43)
  Alopecia: Tumor Assessment Wk 156: number analyzed (Participants) | 8
  Alopecia: Tumor Assessment Wk 156 | -4.17 (45.21)
  Alopecia: Tumor Assessment Wk 165: number analyzed (Participants) | 3
  Alopecia: Tumor Assessment Wk 165 | 0.00 (0.00)
  Alopecia: Tumor Assessment Wk 174: number analyzed (Participants) | 1
  Alopecia: Tumor Assessment Wk 174 | 0.00
  Alopecia: Tumor Assessment Wk 183: number analyzed (Participants) | 1
  Alopecia: Tumor Assessment Wk 183 | 33.33
  Pain in chest: Baseline: number analyzed (Participants) | 582
  Pain in chest: Baseline | 14.20 (21.62)
  Pain in chest: C2D1: number analyzed (Participants) | 497
  Pain in chest: C2D1 | 0.13 (19.74)
  Pain in chest: Tumor Assessment Wk 006: number analyzed (Participants) | 335
  Pain in chest: Tumor Assessment Wk 006 | 0.10 (23.99)
  Pain in chest: Tumor Assessment Wk 012: number analyzed (Participants) | 221
  Pain in chest: Tumor Assessment Wk 012 | -0.75 (22.35)
  Pain in chest: Tumor Assessment Wk 018: number analyzed (Participants) | 178
  Pain in chest: Tumor Assessment Wk 018 | -1.12 (18.38)
  Pain in chest: Tumor Assessment Wk 024: number analyzed (Participants) | 146
  Pain in chest: Tumor Assessment Wk 024 | -2.74 (18.16)
  Pain in chest: Tumor Assessment Wk 030: number analyzed (Participants) | 113
  Pain in chest: Tumor Assessment Wk 030 | -1.77 (20.82)
  Pain in chest: Tumor Assessment Wk 036: number analyzed (Participants) | 90
  Pain in chest: Tumor Assessment Wk 036 | -2.96 (20.39)
  Pain in chest: Tumor Assessment Wk 042: number analyzed (Participants) | 83
  Pain in chest: Tumor Assessment Wk 042 | -2.41 (20.02)
  Pain in chest: Tumor Assessment Wk 048: number analyzed (Participants) | 69
  Pain in chest: Tumor Assessment Wk 048 | -4.35 (22.80)
  Pain in chest: Tumor Assessment Wk 054: number analyzed (Participants) | 12
  Pain in chest: Tumor Assessment Wk 054 | 0.00 (20.10)
  Pain in chest: Tumor Assessment Wk 057: number analyzed (Participants) | 55
  Pain in chest: Tumor Assessment Wk 057 | -6.06 (21.36)
  Pain in chest: Tumor Assessment Wk 060: number analyzed (Participants) | 9
  Pain in chest: Tumor Assessment Wk 060 | 7.41 (22.22)
  Pain in chest: Tumor Assessment Wk 066: number analyzed (Participants) | 50
  Pain in chest: Tumor Assessment Wk 066 | -3.33 (20.48)
  Pain in chest: Tumor Assessment Wk 072: number analyzed (Participants) | 7
  Pain in chest: Tumor Assessment Wk 072 | -14.29 (17.82)
  Pain in chest: Tumor Assessment Wk 075: number analyzed (Participants) | 38
  Pain in chest: Tumor Assessment Wk 075 | -6.14 (18.75)
  Pain in chest: Tumor Assessment Wk 078: number analyzed (Participants) | 4
  Pain in chest: Tumor Assessment Wk 078 | -16.67 (19.25)
  Pain in chest: Tumor Assessment Wk 084: number analyzed (Participants) | 36
  Pain in chest: Tumor Assessment Wk 084 | -7.41 (16.16)
  Pain in chest: Tumor Assessment Wk 090: number analyzed (Participants) | 5
  Pain in chest: Tumor Assessment Wk 090 | -6.67 (14.91)
  Pain in chest: Tumor Assessment Wk 093: number analyzed (Participants) | 25
  Pain in chest: Tumor Assessment Wk 093 | -1.33 (15.15)
  Pain in chest: Tumor Assessment Wk 096: number analyzed (Participants) | 4
  Pain in chest: Tumor Assessment Wk 096 | -8.33 (16.67)
  Pain in chest: Tumor Assessment Wk 102: number analyzed (Participants) | 26
  Pain in chest: Tumor Assessment Wk 102 | -8.97 (15.08)
  Pain in chest: Tumor Assessment Wk 108: number analyzed (Participants) | 5
  Pain in chest: Tumor Assessment Wk 108 | -13.33 (18.26)
  Pain in chest: Tumor Assessment Wk 111: number analyzed (Participants) | 20
  Pain in chest: Tumor Assessment Wk 111 | -5.00 (16.31)
  Pain in chest: Tumor Assessment Wk 114: number analyzed (Participants) | 2
  Pain in chest: Tumor Assessment Wk 114 | -33.33 (0.00)
  Pain in chest: Tumor Assessment Wk 120: number analyzed (Participants) | 18
  Pain in chest: Tumor Assessment Wk 120 | -7.41 (18.28)
  Pain in chest: Tumor Assessment Wk 126: number analyzed (Participants) | 3
  Pain in chest: Tumor Assessment Wk 126 | -11.11 (19.25)
  Pain in chest: Tumor Assessment Wk 129: number analyzed (Participants) | 16
  Pain in chest: Tumor Assessment Wk 129 | -6.25 (18.13)
  Pain in chest: Tumor Assessment Wk 132: number analyzed (Participants) | 1
  Pain in chest: Tumor Assessment Wk 132 | -33.33
  Pain in chest: Tumor Assessment Wk 138: number analyzed (Participants) | 13
  Pain in chest: Tumor Assessment Wk 138 | -5.13 (22.96)
  Pain in chest: Tumor Assessment Wk 144: number analyzed (Participants) | 1
  Pain in chest: Tumor Assessment Wk 144 | -33.33
  Pain in chest: Tumor Assessment Wk 147: number analyzed (Participants) | 8
  Pain in chest: Tumor Assessment Wk 147 | -4.17 (21.36)
  Pain in chest: Tumor Assessment Wk 156: number analyzed (Participants) | 7
  Pain in chest: Tumor Assessment Wk 156 | -9.52 (16.27)
  Pain in chest: Tumor Assessment Wk 165: number analyzed (Participants) | 3
  Pain in chest: Tumor Assessment Wk 165 | 11.11 (19.25)
  Pain in chest: Tumor Assessment Wk 174: number analyzed (Participants) | 1
  Pain in chest: Tumor Assessment Wk 174 | 0.00
  Pain in chest: Tumor Assessment Wk 183: number analyzed (Participants) | 1
  Pain in chest: Tumor Assessment Wk 183 | 33.33
  Pain in arm or shoulder: Baseline: number analyzed (Participants) | 582
  Pain in arm or shoulder: Baseline | 16.09 (24.63)
  Pain in arm or shoulder: C2D1: number analyzed (Participants) | 497
  Pain in arm or shoulder: C2D1 | 1.81 (21.67)
  Pain in arm or shoulder: Tumor Assessment Wk 006: number analyzed (Participants) | 331
  Pain in arm or shoulder: Tumor Assessment Wk 006 | -0.30 (23.85)
  Pain in arm or shoulder: Tumor Assessment Wk 012: number analyzed (Participants) | 221
  Pain in arm or shoulder: Tumor Assessment Wk 012 | 0.75 (24.09)
  Pain in arm or shoulder: Tumor Assessment Wk 018: number analyzed (Participants) | 180
  Pain in arm or shoulder: Tumor Assessment Wk 018 | 3.15 (28.78)
  Pain in arm or shoulder: Tumor Assessment Wk 024: number analyzed (Participants) | 147
  Pain in arm or shoulder: Tumor Assessment Wk 024 | -0.68 (23.56)
  Pain in arm or shoulder: Tumor Assessment Wk 030: number analyzed (Participants) | 114
  Pain in arm or shoulder: Tumor Assessment Wk 030 | 0.00 (25.86)
  Pain in arm or shoulder: Tumor Assessment Wk 036: number analyzed (Participants) | 91
  Pain in arm or shoulder: Tumor Assessment Wk 036 | -2.20 (22.11)
  Pain in arm or shoulder: Tumor Assessment Wk 042: number analyzed (Participants) | 84
  Pain in arm or shoulder: Tumor Assessment Wk 042 | -1.19 (24.51)
  Pain in arm or shoulder: Tumor Assessment Wk 048: number analyzed (Participants) | 70
  Pain in arm or shoulder: Tumor Assessment Wk 048 | -2.38 (24.95)
  Pain in arm or shoulder: Tumor Assessment Wk 054: number analyzed (Participants) | 13
  Pain in arm or shoulder: Tumor Assessment Wk 054 | 2.56 (21.35)
  Pain in arm or shoulder: Tumor Assessment Wk 057: number analyzed (Participants) | 58
  Pain in arm or shoulder: Tumor Assessment Wk 057 | 1.72 (26.80)
  Pain in arm or shoulder: Tumor Assessment Wk 060: number analyzed (Participants) | 10
  Pain in arm or shoulder: Tumor Assessment Wk 060 | -6.67 (21.08)
  Pain in arm or shoulder: Tumor Assessment Wk 066: number analyzed (Participants) | 52
  Pain in arm or shoulder: Tumor Assessment Wk 066 | 0.64 (21.38)
  Pain in arm or shoulder: Tumor Assessment Wk 072: number analyzed (Participants) | 7
  Pain in arm or shoulder: Tumor Assessment Wk 072 | 4.76 (23.00)
  Pain in arm or shoulder: Tumor Assessment Wk 075: number analyzed (Participants) | 39
  Pain in arm or shoulder: Tumor Assessment Wk 075 | -4.27 (23.17)
  Pain in arm or shoulder: Tumor Assessment Wk 078: number analyzed (Participants) | 4
  Pain in arm or shoulder: Tumor Assessment Wk 078 | 16.67 (19.25)
  Pain in arm or shoulder: Tumor Assessment Wk 084: number analyzed (Participants) | 37
  Pain in arm or shoulder: Tumor Assessment Wk 084 | -9.01 (23.11)
  Pain in arm or shoulder: Tumor Assessment Wk 090: number analyzed (Participants) | 5
  Pain in arm or shoulder: Tumor Assessment Wk 090 | 0.00 (23.57)
  Pain in arm or shoulder: Tumor Assessment Wk 093: number analyzed (Participants) | 27
  Pain in arm or shoulder: Tumor Assessment Wk 093 | -9.88 (20.29)
  Pain in arm or shoulder: Tumor Assessment Wk 096: number analyzed (Participants) | 4
  Pain in arm or shoulder: Tumor Assessment Wk 096 | -8.33 (16.67)
  Pain in arm or shoulder: Tumor Assessment Wk 102: number analyzed (Participants) | 27
  Pain in arm or shoulder: Tumor Assessment Wk 102 | -4.94 (20.05)
  Pain in arm or shoulder: Tumor Assessment Wk 108: number analyzed (Participants) | 5
  Pain in arm or shoulder: Tumor Assessment Wk 108 | 0.00 (23.57)
  Pain in arm or shoulder: Tumor Assessment Wk 111: number analyzed (Participants) | 21
  Pain in arm or shoulder: Tumor Assessment Wk 111 | -6.35 (20.05)
  Pain in arm or shoulder: Tumor Assessment Wk 114: number analyzed (Participants) | 2
  Pain in arm or shoulder: Tumor Assessment Wk 114 | 16.67 (23.57)
  Pain in arm or shoulder: Tumor Assessment Wk 120: number analyzed (Participants) | 19
  Pain in arm or shoulder: Tumor Assessment Wk 120 | -7.02 (21.02)
  Pain in arm or shoulder: Tumor Assessment Wk 126: number analyzed (Participants) | 3
  Pain in arm or shoulder: Tumor Assessment Wk 126 | 22.22 (19.25)
  Pain in arm or shoulder: Tumor Assessment Wk 129: number analyzed (Participants) | 17
  Pain in arm or shoulder: Tumor Assessment Wk 129 | -7.84 (18.74)
  Pain in arm or shoulder: Tumor Assessment Wk 132: number analyzed (Participants) | 1
  Pain in arm or shoulder: Tumor Assessment Wk 132 | 0.00
  Pain in arm or shoulder: Tumor Assessment Wk 138: number analyzed (Participants) | 14
  Pain in arm or shoulder: Tumor Assessment Wk 138 | -11.90 (16.57)
  Pain in arm or shoulder: Tumor Assessment Wk 144: number analyzed (Participants) | 1
  Pain in arm or shoulder: Tumor Assessment Wk 144 | -33.33
  Pain in arm or shoulder: Tumor Assessment Wk 147: number analyzed (Participants) | 9
  Pain in arm or shoulder: Tumor Assessment Wk 147 | -11.11 (16.67)
  Pain in arm or shoulder: Tumor Assessment Wk 156: number analyzed (Participants) | 8
  Pain in arm or shoulder: Tumor Assessment Wk 156 | -12.50 (17.25)
  Pain in arm or shoulder: Tumor Assessment Wk 165: number analyzed (Participants) | 3
  Pain in arm or shoulder: Tumor Assessment Wk 165 | -11.11 (19.25)
  Pain in arm or shoulder: Tumor Assessment Wk 174: number analyzed (Participants) | 1
  Pain in arm or shoulder: Tumor Assessment Wk 174 | -33.33
  Pain in arm or shoulder: Tumor Assessment Wk 183: number analyzed (Participants) | 1
  Pain in arm or shoulder: Tumor Assessment Wk 183 | 0.00
  Pain in other parts: Baseline: number analyzed (Participants) | 576
  Pain in other parts: Baseline | 25.46 (30.26)
  Pain in other parts: C2D1: number analyzed (Participants) | 481
  Pain in other parts: C2D1 | -0.49 (27.84)
  Pain in other parts: Tumor Assessment Wk 006: number analyzed (Participants) | 327
  Pain in other parts: Tumor Assessment Wk 006 | 1.12 (31.80)
  Pain in other parts: Tumor Assessment Wk 012: number analyzed (Participants) | 214
  Pain in other parts: Tumor Assessment Wk 012 | 0.93 (28.33)
  Pain in other parts: Tumor Assessment Wk 018: number analyzed (Participants) | 168
  Pain in other parts: Tumor Assessment Wk 018 | -1.19 (23.89)
  Pain in other parts: Tumor Assessment Wk 024: number analyzed (Participants) | 142
  Pain in other parts: Tumor Assessment Wk 024 | -1.41 (23.11)
  Pain in other parts: Tumor Assessment Wk 030: number analyzed (Participants) | 107
  Pain in other parts: Tumor Assessment Wk 030 | -0.62 (21.95)
  Pain in other parts: Tumor Assessment Wk 036: number analyzed (Participants) | 88
  Pain in other parts: Tumor Assessment Wk 036 | -4.17 (19.45)
  Pain in other parts: Tumor Assessment Wk 042: number analyzed (Participants) | 80
  Pain in other parts: Tumor Assessment Wk 042 | -4.17 (24.52)
  Pain in other parts: Tumor Assessment Wk 048: number analyzed (Participants) | 68
  Pain in other parts: Tumor Assessment Wk 048 | -0.98 (23.72)
  Pain in other parts: Tumor Assessment Wk 054: number analyzed (Participants) | 12
  Pain in other parts: Tumor Assessment Wk 054 | 11.11 (16.41)
  Pain in other parts: Tumor Assessment Wk 057: number analyzed (Participants) | 51
  Pain in other parts: Tumor Assessment Wk 057 | -5.23 (20.41)
  Pain in other parts: Tumor Assessment Wk 060: number analyzed (Participants) | 9
  Pain in other parts: Tumor Assessment Wk 060 | 3.70 (11.11)
  Pain in other parts: Tumor Assessment Wk 066: number analyzed (Participants) | 50
  Pain in other parts: Tumor Assessment Wk 066 | -0.67 (27.35)
  Pain in other parts: Tumor Assessment Wk 072: number analyzed (Participants) | 7
  Pain in other parts: Tumor Assessment Wk 072 | 4.76 (12.60)
  Pain in other parts: Tumor Assessment Wk 075: number analyzed (Participants) | 37
  Pain in other parts: Tumor Assessment Wk 075 | -2.70 (25.31)
  Pain in other parts: Tumor Assessment Wk 078: number analyzed (Participants) | 4
  Pain in other parts: Tumor Assessment Wk 078 | 16.67 (19.25)
  Pain in other parts: Tumor Assessment Wk 084: number analyzed (Participants) | 34
  Pain in other parts: Tumor Assessment Wk 084 | -3.92 (26.92)
  Pain in other parts: Tumor Assessment Wk 090: number analyzed (Participants) | 5
  Pain in other parts: Tumor Assessment Wk 090 | 6.67 (14.91)
  Pain in other parts: Tumor Assessment Wk 093: number analyzed (Participants) | 26
  Pain in other parts: Tumor Assessment Wk 093 | -10.26 (22.65)
  Pain in other parts: Tumor Assessment Wk 096: number analyzed (Participants) | 3
  Pain in other parts: Tumor Assessment Wk 096 | 0.00 (0.00)
  Pain in other parts: Tumor Assessment Wk 102: number analyzed (Participants) | 26
  Pain in other parts: Tumor Assessment Wk 102 | -8.97 (22.23)
  Pain in other parts: Tumor Assessment Wk 108: number analyzed (Participants) | 5
  Pain in other parts: Tumor Assessment Wk 108 | 6.67 (14.91)
  Pain in other parts: Tumor Assessment Wk 111: number analyzed (Participants) | 20
  Pain in other parts: Tumor Assessment Wk 111 | -8.33 (28.36)
  Pain in other parts: Tumor Assessment Wk 114: number analyzed (Participants) | 2
  Pain in other parts: Tumor Assessment Wk 114 | 16.67 (23.57)
  Pain in other parts: Tumor Assessment Wk 120: number analyzed (Participants) | 17
  Pain in other parts: Tumor Assessment Wk 120 | -3.92 (20.01)
  Pain in other parts: Tumor Assessment Wk 126: number analyzed (Participants) | 3
  Pain in other parts: Tumor Assessment Wk 126 | 33.33 (33.33)
  Pain in other parts: Tumor Assessment Wk 129: number analyzed (Participants) | 16
  Pain in other parts: Tumor Assessment Wk 129 | -6.25 (18.13)
  Pain in other parts: Tumor Assessment Wk 132: number analyzed (Participants) | 1
  Pain in other parts: Tumor Assessment Wk 132 | 0.00
  Pain in other parts: Tumor Assessment Wk 138: number analyzed (Participants) | 13
  Pain in other parts: Tumor Assessment Wk 138 | -10.26 (21.01)
  Pain in other parts: Tumor Assessment Wk 144: number analyzed (Participants) | 1
  Pain in other parts: Tumor Assessment Wk 144 | 0.00
  Pain in other parts: Tumor Assessment Wk 147: number analyzed (Participants) | 8
  Pain in other parts: Tumor Assessment Wk 147 | -12.50 (24.80)
  Pain in other parts: Tumor Assessment Wk 156: number analyzed (Participants) | 7
  Pain in other parts: Tumor Assessment Wk 156 | -14.29 (17.82)
  Pain in other parts: Tumor Assessment Wk 165: number analyzed (Participants) | 3
  Pain in other parts: Tumor Assessment Wk 165 | 0.00 (0.00)
  Pain in other parts: Tumor Assessment Wk 174: number analyzed (Participants) | 1
  Pain in other parts: Tumor Assessment Wk 174 | 0.00
  Pain in other parts: Tumor Assessment Wk 183: number analyzed (Participants) | 1
  Pain in other parts: Tumor Assessment Wk 183 | 0.00
  Dyspnoea at Resting: Baseline: number analyzed (Participants) | 586
  Dyspnoea at Resting: Baseline | 10.47 (19.79)
  Dyspnoea at Resting: C2D1: number analyzed (Participants) | 500
  Dyspnoea at Resting: C2D1 | 2.53 (19.17)
  Dyspnoea at Resting: Tumor Assessment Wk 006: number analyzed (Participants) | 337
  Dyspnoea at Resting: Tumor Assessment Wk 006 | 1.68 (20.59)
  Dyspnoea at Resting: Tumor Assessment Wk 012: number analyzed (Participants) | 222
  Dyspnoea at Resting: Tumor Assessment Wk 012 | 1.65 (19.61)
  Dyspnoea at Resting: Tumor Assessment Wk 018: number analyzed (Participants) | 182
  Dyspnoea at Resting: Tumor Assessment Wk 018 | 1.83 (17.07)
  Dyspnoea at Resting: Tumor Assessment Wk 024: number analyzed (Participants) | 146
  Dyspnoea at Resting: Tumor Assessment Wk 024 | -0.23 (15.90)
  Dyspnoea at Resting: Tumor Assessment Wk 030: number analyzed (Participants) | 115
  Dyspnoea at Resting: Tumor Assessment Wk 030 | 2.03 (21.76)
  Dyspnoea at Resting: Tumor Assessment Wk 036: number analyzed (Participants) | 91
  Dyspnoea at Resting: Tumor Assessment Wk 036 | 0.37 (20.18)
  Dyspnoea at Resting: Tumor Assessment Wk 042: number analyzed (Participants) | 84
  Dyspnoea at Resting: Tumor Assessment Wk 042 | -0.40 (19.01)
  Dyspnoea at Resting: Tumor Assessment Wk 048: number analyzed (Participants) | 70
  Dyspnoea at Resting: Tumor Assessment Wk 048 | 0.95 (17.92)
  Dyspnoea at Resting: Tumor Assessment Wk 054: number analyzed (Participants) | 14
  Dyspnoea at Resting: Tumor Assessment Wk 054 | 2.38 (8.91)
  Dyspnoea at Resting: Tumor Assessment Wk 057: number analyzed (Participants) | 56
  Dyspnoea at Resting: Tumor Assessment Wk 057 | -2.38 (19.96)
  Dyspnoea at Resting: Tumor Assessment Wk 060: number analyzed (Participants) | 10
  Dyspnoea at Resting: Tumor Assessment Wk 060 | 0.00 (0.00)
  Dyspnoea at Resting: Tumor Assessment Wk 066: number analyzed (Participants) | 51
  Dyspnoea at Resting: Tumor Assessment Wk 066 | 3.27 (17.96)
  Dyspnoea at Resting: Tumor Assessment Wk 072: number analyzed (Participants) | 7
  Dyspnoea at Resting: Tumor Assessment Wk 072 | 9.52 (31.71)
  Dyspnoea at Resting: Tumor Assessment Wk 075: number analyzed (Participants) | 40
  Dyspnoea at Resting: Tumor Assessment Wk 075 | -0.83 (17.68)
  Dyspnoea at Resting: Tumor Assessment Wk 078: number analyzed (Participants) | 5
  Dyspnoea at Resting: Tumor Assessment Wk 078 | 20.00 (50.55)
  Dyspnoea at Resting: Tumor Assessment Wk 084: number analyzed (Participants) | 38
  Dyspnoea at Resting: Tumor Assessment Wk 084 | -0.88 (16.42)
  Dyspnoea at Resting: Tumor Assessment Wk 090: number analyzed (Participants) | 6
  Dyspnoea at Resting: Tumor Assessment Wk 090 | 11.11 (45.54)
  Dyspnoea at Resting: Tumor Assessment Wk 093: number analyzed (Participants) | 28
  Dyspnoea at Resting: Tumor Assessment Wk 093 | 4.76 (23.51)
  Dyspnoea at Resting: Tumor Assessment Wk 096: number analyzed (Participants) | 5
  Dyspnoea at Resting: Tumor Assessment Wk 096 | 13.33 (29.81)
  Dyspnoea at Resting: Tumor Assessment Wk 102: number analyzed (Participants) | 28
  Dyspnoea at Resting: Tumor Assessment Wk 102 | -1.19 (16.93)
  Dyspnoea at Resting: Tumor Assessment Wk 108: number analyzed (Participants) | 5
  Dyspnoea at Resting: Tumor Assessment Wk 108 | -6.67 (27.89)
  Dyspnoea at Resting: Tumor Assessment Wk 111: number analyzed (Participants) | 21
  Dyspnoea at Resting: Tumor Assessment Wk 111 | -1.59 (16.59)
  Dyspnoea at Resting: Tumor Assessment Wk 114: number analyzed (Participants) | 2
  Dyspnoea at Resting: Tumor Assessment Wk 114 | -16.67 (23.57)
  Dyspnoea at Resting: Tumor Assessment Wk 120: number analyzed (Participants) | 19
  Dyspnoea at Resting: Tumor Assessment Wk 120 | -1.75 (13.49)
  Dyspnoea at Resting: Tumor Assessment Wk 126: number analyzed (Participants) | 3
  Dyspnoea at Resting: Tumor Assessment Wk 126 | -11.11 (19.25)
  Dyspnoea at Resting: Tumor Assessment Wk 129: number analyzed (Participants) | 17
  Dyspnoea at Resting: Tumor Assessment Wk 129 | -1.96 (14.29)
  Dyspnoea at Resting: Tumor Assessment Wk 132: number analyzed (Participants) | 1
  Dyspnoea at Resting: Tumor Assessment Wk 132 | 0.00
  Dyspnoea at Resting: Tumor Assessment Wk 138: number analyzed (Participants) | 13
  Dyspnoea at Resting: Tumor Assessment Wk 138 | 7.69 (19.97)
  Dyspnoea at Resting: Tumor Assessment Wk 144: number analyzed (Participants) | 1
  Dyspnoea at Resting: Tumor Assessment Wk 144 | 0.00
  Dyspnoea at Resting: Tumor Assessment Wk 147: number analyzed (Participants) | 9
  Dyspnoea at Resting: Tumor Assessment Wk 147 | 7.41 (14.70)
  Dyspnoea at Resting: Tumor Assessment Wk 156: number analyzed (Participants) | 8
  Dyspnoea at Resting: Tumor Assessment Wk 156 | 20.83 (17.25)
  Dyspnoea at Resting: Tumor Assessment Wk 165: number analyzed (Participants) | 3
  Dyspnoea at Resting: Tumor Assessment Wk 165 | 11.11 (19.25)
  Dyspnoea at Resting: Tumor Assessment Wk 174: number analyzed (Participants) | 1
  Dyspnoea at Resting: Tumor Assessment Wk 174 | 0.00
  Dyspnoea at Resting: Tumor Assessment Wk 183: number analyzed (Participants) | 1
  Dyspnoea at Resting: Tumor Assessment Wk 183 | 33.33
  Dyspnoea at Walking: Baseline: number analyzed (Participants) | 587
  Dyspnoea at Walking: Baseline | 27.31 (26.59)
  Dyspnoea at Walking: C2D1: number analyzed (Participants) | 502
  Dyspnoea at Walking: C2D1 | 2.52 (21.43)
  Dyspnoea at Walking: Tumor Assessment Wk 006: number analyzed (Participants) | 338
  Dyspnoea at Walking: Tumor Assessment Wk 006 | 1.18 (23.65)
  Dyspnoea at Walking: Tumor Assessment Wk 012: number analyzed (Participants) | 221
  Dyspnoea at Walking: Tumor Assessment Wk 012 | -1.21 (26.37)
  Dyspnoea at Walking: Tumor Assessment Wk 018: number analyzed (Participants) | 181
  Dyspnoea at Walking: Tumor Assessment Wk 018 | -1.29 (24.94)
  Dyspnoea at Walking: Tumor Assessment Wk 024: number analyzed (Participants) | 148
  Dyspnoea at Walking: Tumor Assessment Wk 024 | -3.83 (26.23)
  Dyspnoea at Walking: Tumor Assessment Wk 030: number analyzed (Participants) | 115
  Dyspnoea at Walking: Tumor Assessment Wk 030 | -2.32 (26.39)
  Dyspnoea at Walking: Tumor Assessment Wk 036: number analyzed (Participants) | 93
  Dyspnoea at Walking: Tumor Assessment Wk 036 | -3.94 (27.74)
  Dyspnoea at Walking: Tumor Assessment Wk 042: number analyzed (Participants) | 86
  Dyspnoea at Walking: Tumor Assessment Wk 042 | -3.88 (25.78)
  Dyspnoea at Walking: Tumor Assessment Wk 048: number analyzed (Participants) | 72
  Dyspnoea at Walking: Tumor Assessment Wk 048 | -6.48 (27.77)
  Dyspnoea at Walking: Tumor Assessment Wk 054: number analyzed (Participants) | 14
  Dyspnoea at Walking: Tumor Assessment Wk 054 | 2.38 (27.62)
  Dyspnoea at Walking: Tumor Assessment Wk 057: number analyzed (Participants) | 57
  Dyspnoea at Walking: Tumor Assessment Wk 057 | -7.02 (23.35)
  Dyspnoea at Walking: Tumor Assessment Wk 060: number analyzed (Participants) | 11
  Dyspnoea at Walking: Tumor Assessment Wk 060 | -3.03 (17.98)
  Dyspnoea at Walking: Tumor Assessment Wk 066: number analyzed (Participants) | 53
  Dyspnoea at Walking: Tumor Assessment Wk 066 | -1.89 (25.67)
  Dyspnoea at Walking: Tumor Assessment Wk 072: number analyzed (Participants) | 7
  Dyspnoea at Walking: Tumor Assessment Wk 072 | 4.76 (29.99)
  Dyspnoea at Walking: Tumor Assessment Wk 075: number analyzed (Participants) | 40
  Dyspnoea at Walking: Tumor Assessment Wk 075 | -4.17 (22.88)
  Dyspnoea at Walking: Tumor Assessment Wk 078: number analyzed (Participants) | 5
  Dyspnoea at Walking: Tumor Assessment Wk 078 | -6.67 (54.77)
  Dyspnoea at Walking: Tumor Assessment Wk 084: number analyzed (Participants) | 38
  Dyspnoea at Walking: Tumor Assessment Wk 084 | -6.14 (23.06)
  Dyspnoea at Walking: Tumor Assessment Wk 090: number analyzed (Participants) | 6
  Dyspnoea at Walking: Tumor Assessment Wk 090 | -5.56 (38.97)
  Dyspnoea at Walking: Tumor Assessment Wk 093: number analyzed (Participants) | 28
  Dyspnoea at Walking: Tumor Assessment Wk 093 | -5.95 (24.09)
  Dyspnoea at Walking: Tumor Assessment Wk 096: number analyzed (Participants) | 5
  Dyspnoea at Walking: Tumor Assessment Wk 096 | 13.33 (38.01)
  Dyspnoea at Walking: Tumor Assessment Wk 102: number analyzed (Participants) | 28
  Dyspnoea at Walking: Tumor Assessment Wk 102 | -8.33 (26.64)
  Dyspnoea at Walking: Tumor Assessment Wk 108: number analyzed (Participants) | 5
  Dyspnoea at Walking: Tumor Assessment Wk 108 | -20.00 (29.81)
  Dyspnoea at Walking: Tumor Assessment Wk 111: number analyzed (Participants) | 21
  Dyspnoea at Walking: Tumor Assessment Wk 111 | -9.52 (26.13)
  Dyspnoea at Walking: Tumor Assessment Wk 114: number analyzed (Participants) | 2
  Dyspnoea at Walking: Tumor Assessment Wk 114 | -16.67 (23.57)
  Dyspnoea at Walking: Tumor Assessment Wk 120: number analyzed (Participants) | 19
  Dyspnoea at Walking: Tumor Assessment Wk 120 | -7.02 (21.02)
  Dyspnoea at Walking: Tumor Assessment Wk 126: number analyzed (Participants) | 3
  Dyspnoea at Walking: Tumor Assessment Wk 126 | -33.33 (33.33)
  Dyspnoea at Walking: Tumor Assessment Wk 129: number analyzed (Participants) | 17
  Dyspnoea at Walking: Tumor Assessment Wk 129 | -9.80 (19.60)
  Dyspnoea at Walking: Tumor Assessment Wk 132: number analyzed (Participants) | 1
  Dyspnoea at Walking: Tumor Assessment Wk 132 | -33.33
  Dyspnoea at Walking: Tumor Assessment Wk 138: number analyzed (Participants) | 14
  Dyspnoea at Walking: Tumor Assessment Wk 138 | -2.38 (24.33)
  Dyspnoea at Walking: Tumor Assessment Wk 144: number analyzed (Participants) | 1
  Dyspnoea at Walking: Tumor Assessment Wk 144 | 0.00
  Dyspnoea at Walking: Tumor Assessment Wk 147: number analyzed (Participants) | 9
  Dyspnoea at Walking: Tumor Assessment Wk 147 | -3.70 (26.06)
  Dyspnoea at Walking: Tumor Assessment Wk 156: number analyzed (Participants) | 8
  Dyspnoea at Walking: Tumor Assessment Wk 156 | 4.17 (37.53)
  Dyspnoea at Walking: Tumor Assessment Wk 165: number analyzed (Participants) | 3
  Dyspnoea at Walking: Tumor Assessment Wk 165 | 11.11 (38.49)
  Dyspnoea at Walking: Tumor Assessment Wk 174: number analyzed (Participants) | 1
  Dyspnoea at Walking: Tumor Assessment Wk 174 | 0.00
  Dyspnoea at Walking: Tumor Assessment Wk 183: number analyzed (Participants) | 1
  Dyspnoea at Walking: Tumor Assessment Wk 183 | -33.33
  Dyspnoea at Climbing Stairs: Baseline: number analyzed (Participants) | 581
  Dyspnoea at Climbing Stairs: Baseline | 37.12 (29.57)
  Dyspnoea at Climbing Stairs: C2D1: number analyzed (Participants) | 494
  Dyspnoea at Climbing Stairs: C2D1 | 2.23 (22.71)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 006: number analyzed (Participants) | 336
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 006 | 1.39 (26.23)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 012: number analyzed (Participants) | 221
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 012 | -1.66 (27.20)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 018: number analyzed (Participants) | 180
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 018 | -2.04 (26.17)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 024: number analyzed (Participants) | 148
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 024 | -4.73 (24.90)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 030: number analyzed (Participants) | 115
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 030 | -2.61 (28.66)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 036: number analyzed (Participants) | 93
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 036 | -6.81 (29.72)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 042: number analyzed (Participants) | 86
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 042 | -5.81 (26.17)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 048: number analyzed (Participants) | 72
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 048 | -3.70 (29.37)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 054: number analyzed (Participants) | 14
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 054 | 2.38 (24.33)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 057: number analyzed (Participants) | 58
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 057 | -6.90 (27.75)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 060: number analyzed (Participants) | 11
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 060 | -3.03 (17.98)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 066: number analyzed (Participants) | 53
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 066 | 1.89 (26.49)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 072: number analyzed (Participants) | 7
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 072 | 0.00 (33.33)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 075: number analyzed (Participants) | 40
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 075 | -1.67 (28.19)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 078: number analyzed (Participants) | 5
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 078 | -13.33 (29.81)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 084: number analyzed (Participants) | 38
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 084 | -1.75 (24.44)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 090: number analyzed (Participants) | 5
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 090 | -26.67 (14.91)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 093: number analyzed (Participants) | 28
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 093 | -9.52 (23.76)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 096: number analyzed (Participants) | 5
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 096 | 13.33 (29.81)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 102: number analyzed (Participants) | 28
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 102 | -8.33 (26.64)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 108: number analyzed (Participants) | 5
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 108 | 0.00 (33.33)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 111: number analyzed (Participants) | 21
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 111 | -9.52 (23.90)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 114: number analyzed (Participants) | 2
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 114 | -16.67 (23.57)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 120: number analyzed (Participants) | 19
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 120 | -8.77 (18.73)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 126: number analyzed (Participants) | 3
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 126 | -11.11 (38.49)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 129: number analyzed (Participants) | 17
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 129 | -9.80 (22.87)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 132: number analyzed (Participants) | 1
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 132 | -33.33
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 138: number analyzed (Participants) | 14
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 138 | -11.90 (24.83)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 144: number analyzed (Participants) | 1
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 144 | 0.00
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 147: number analyzed (Participants) | 9
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 147 | -14.81 (17.57)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 156: number analyzed (Participants) | 8
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 156 | -4.17 (27.82)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 165: number analyzed (Participants) | 3
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 165 | -11.11 (19.25)
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 174: number analyzed (Participants) | 1
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 174 | 0.00
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 183: number analyzed (Participants) | 1
  Dyspnoea at Climbing Stairs: Tumor Assessment Wk 183 | -33.33

12. Secondary Outcome: Progression-Free Survival as Evaluated By the Investigator in Accordance With Modified RECIST
Description: PFS was defined as the time (in months) from initiation of study treatment to the first documented disease progression or death from any cause, whichever occurred first. PFS was evaluated by the investigator according to modified RECIST.
Time Frame: Baseline up to disease progression or death whichever occurs first (up to 4 years)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Months | 3.7 [3.0 to 4.2]

13. Secondary Outcome: Percentage of Participants Alive 3 Years After Initiation of Treatment
Description: The OS rate at 3 years, was defined as the percentage of participants remaining alive 3 years after initiation of study treatment.
Time Frame: Baseline up to Year 3
Population: The safety population was based on all participants who received any dose of atezolizumab during the study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Percentage of Participants | 19.6

14. Secondary Outcome: Percentage of Participants With Objective Reponse as Assessed by the Investigator According to RECIST v1.1
Description: Objective response rate (ORR), according to RECIST v1.1, was defined as the percentage of participants with a confirmed best overall response (BOR), either complete response (CR) or partial response (PR), as determined by the investigator using RECIST v1.1.
Time Frame: Baseline up to disease progression or death whichever occurs first (up to 4 years)
Population: The safety population was based on all participants who received any dose of atezolizumab during the study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Percentage of Participants | 11.5

15. Secondary Outcome: Percentage of Participants With Objective Reponse as Assessed by the Investigator According to Modified RECIST
Description: The investigator-assessed ORR was defined as the proportion of participants whose confirmed BOR is either a PR or CR per modified RECIST.
Time Frame: Baseline up to disease progression or death whichever occurs first (up to 4 years)
Population: The safety population was based on all participants who received any dose of atezolizumab during the study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Percentage of Participants | 12.4

16. Secondary Outcome: Duration of Response as Assessed by the Investigator According to RECIST v.1.1
Description: DOR was defined as the time from the first tumor assessment that supported the participant's objective response (CR or PR, whichever was first reported) to documented disease progression as determined by the investigator according to RECIST v1.1 or death from any cause, whichever occurred first, among participants who had a best overall response as CR or PR.
Time Frame: From date of first objective response up to disease progression or death whichever occurs first (up to 4 years)
Population: The safety population was based on all participants who received any dose of atezolizumab during the study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Months | 16.6 [9.7 to 20.3]

17. Secondary Outcome: Duration of Response as Assessed by the Investigator According to Modified RECIST
Description: DOR was defined as the duration from the first tumor assessment that supports the participant's objective response (CR or PR, whichever is first recorded) to disease progression or death due to any cause, whichever occurred first.
Time Frame: From date of first objective response up to disease progression or death whichever occurs first (up to 4 years)
Population: The safety population was based on all participants who received any dose of atezolizumab during the study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 615
Months | 20.5 [16.6 to 28.8]

ADVERSE EVENTS:
Time Frame: Baseline up to 4 years
Description: The ITT population consisted of 619 enrolled participants and the safety population consisted of the 615 participants who received at least one dose of atezolizumab, which was the primary analysis population for the study. Four enrolled participants died before receiving the treatment and were excluded from the safety population. They are included in the all-cause mortality count.
Arm/Group | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 474/619
Serious Adverse Events (participants affected / at risk) | 198/615
Other Adverse Events (participants affected / at risk) | 480/615
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=615)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (2)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 4 (4)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2)
Endocarditis noninfective (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 4 (4)
Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Primary adrenal insufficiency (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Chest pain (General disorders) | 2 (2)
Death (General disorders) | 2 (2)
Device related thrombosis (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 2 (2)
Influenza like illness (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 7 (8)
Sudden death (General disorders) | 2 (2)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Anaphylactic shock (Immune system disorders) | 2 (2)
Atypical pneumonia (Infections and infestations) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Diverticulitis (Infections and infestations) | 2 (2)
Encephalitis (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (2)
Erysipelas (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Infected fistula (Infections and infestations) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 11 (12)
Pleural infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 35 (39)
Pneumonia bacterial (Infections and infestations) | 2 (2)
Pneumonia escherichia (Infections and infestations) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (5)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal cord injury (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 2 (2)
Epilepsy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2)
Neurological symptom (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (2)
Syncope (Nervous system disorders) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Limb operation (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Embolism venous (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Jugular vein thrombosis (Vascular disorders) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=615)
Anaemia (Blood and lymphatic system disorders) | 78 (99)
Hyperthyroidism (Endocrine disorders) | 42 (50)
Hypothyroidism (Endocrine disorders) | 62 (87)
Constipation (Gastrointestinal disorders) | 55 (68)
Diarrhoea (Gastrointestinal disorders) | 72 (97)
Nausea (Gastrointestinal disorders) | 67 (89)
Vomiting (Gastrointestinal disorders) | 46 (59)
Asthenia (General disorders) | 93 (123)
Fatigue (General disorders) | 100 (111)
Pyrexia (General disorders) | 73 (123)
Nasopharyngitis (Infections and infestations) | 35 (44)
Upper respiratory tract infection (Infections and infestations) | 36 (44)
Urinary tract infection (Infections and infestations) | 43 (60)
Decreased appetite (Metabolism and nutrition disorders) | 104 (116)
Hyperglycaemia (Metabolism and nutrition disorders) | 33 (40)
Arthralgia (Musculoskeletal and connective tissue disorders) | 83 (102)
Back pain (Musculoskeletal and connective tissue disorders) | 63 (76)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 37 (39)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 39 (45)
Headache (Nervous system disorders) | 44 (47)
Cough (Respiratory, thoracic and mediastinal disorders) | 107 (134)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 85 (97)
Pruritus (Skin and subcutaneous tissue disorders) | 46 (55)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT03285763/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT03285763/SAP_001.pdf